- 16.1.9 **Documentation of Statistical Methods**
- 16.1.9.1 Statistical Analysis Plan



## STATISTICAL ANALYSIS PLAN

A single-center, randomized, controlled, open-label study in smoking healthy subjects to investigate the nicotine pharmacokinetic profiles following single use of Tobacco Heating System (THS) with a regular or a menthol stick, compared to smoking of a single combustible cigarette (CIG)

Short Title: Nicotine pharmacokinetics of THS single use of a regular or a menthol stick compared to CIG

Protocol No: P1-PK-12 Protocol Version 1.0 Date: 22 November 2022 Protocol Version 2.0 (Protocol Amendment) Date: 06 February 2023

Test Product Name: Tobacco Heating System (THS) Induction device and regular or menthol sticks

Project CA39924 Final Version 1.0 Date: 15 March 2023

Philip Morris Products S.A. Quai Jeanrenaud 3 2000 Neuchâtel, Switzerland



THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

#### STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Test Product Name: Tobacco Heating System (THS) Induction device and regular or menthol sticks

Protocol: P1-PK-12

Study Title: A single-center, randomized, controlled, open-label study in smoking healthy subjects to investigate the nicotine pharmacokinetic profiles following single use of Tobacco Heating System (THS) with a regular or a menthol stick, compared to smoking of a single combustible cigarette (CIG)

Short Title: Nicotine pharmacokinetics of THS single use of a regular or a menthol stick compared to CIG

Issue Date: 15 March 2023



# THS Induction device and regular or menthol sticks, P1-PK-12

# CA39924

# **TABLE OF CONTENTS**

| STA | ATIST | ΓICAL ANALYSIS PLAN | 1 |
|---|---|---|---|
| STA | ATIS | ΓΙCAL ANALYSIS PLAN SIGNATURE PAGE | 2 |
| TA | BLE ( | OF CONTENTS | 3 |
| 1. | INT | RODUCTION | 5 |
| 2. | | ECTIVES AND ENDPOINTS | |
| 3. | | DY DESIGN | |
| 4. | 4.1 | ALYSIS POPULATIONS | |
| | 4.1 | Safety Population (SAF) | |
| | 4.2 | Randomized Population | |
| | 4.4 | Pharmacokinetic Population. | |
| | 7.7 | 4.4.1 Protocol Deviations | |
| 5. | PRO | DUCT DESCRIPTIONS | |
| J. | 5.1 | Test Products | |
| | 5.2 | Comparator Product | |
| 6. | | RMACOKINETIC ANALYSIS | |
| 0. | 6.1 | Collection Schedule for Plasma Nicotine | |
| | 6.2 | Plasma Nicotine Concentrations | |
| | 6.3 | Plasma Nicotine Pharmacokinetic Parameters | |
| | 6.4 | Data Summarization and Presentation | |
| | 6.5 | Statistical Analysis of Pharmacokinetic Parameters | |
| | | 6.5.1 Main Analysis | 13 |
| | | 6.5.2 Sensitivity Analyses | 14 |
| | | 6.5.3 Supplementary Analysis | 14 |
| | 6.6 | Preliminary Data and Interim Analysis | 14 |
| 7. | PHA | RMACODYNAMIC EFFECTS (SUBJECTIVE EFFECTS) | 14 |
| | 7.1 | Data Collection | 14 |
| | 7.2 | Data Summarization. | 14 |
| 8. | SAF | ETY | 15 |
| | 8.1 | Subject Disposition | 15 |
| | 8.2 | Protocol Deviations | 15 |
| | 8.3 | Demographics | 16 |
| | 8.4 | Tobacco/Nicotine-Containing Product Use History Questionnaire | 16 |
| | 8.5 | Usual Brand Cigarettes Documentation. | 16 |

# THS Induction device and regular or menthol sticks, P1-PK-12

# CA39924

| | 8.6 | Fagerström Test for Nicotine Dependence (FTND) | |
|---|---|---|---|
| | 8.7 | Medical History. | 17 |
| | 8.8 | Adverse Events | 17 |
| | 8.9 | Clinical Laboratory Tests (Serum Chemistry, Hematology, and Urinalysis) | 17 |
| | 8.10 | Vital Signs | 18 |
| | 8.11 | Electrocardiogram | 19 |
| | 8.12 | Prior and Concomitant Medications and Concomitant Procedures | 19 |
| | 8.13 | Physical Examination | 19 |
| | 8.14 | Spirometry | 19 |
| | 8.15 | Product Events | 20 |
| 9. | SUM | MARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 20 |
| 10. | REFI | ERENCES | 20 |
| 11. | SUM | MARY TABLES, FIGURES, AND LISTINGS | 21 |
| | 11.1 | In-text Summary Tables and Figures | 21 |
| | 11.2 | Section 14 Summary Tables and Figures | 22 |
| | 11.3 | Section 16 Data Listings | 26 |
| 12. | TAB | LE, FIGURE, AND LISTING SHELLS | 29 |
| | 12.1 | In-text Summary Tables Shells | 30 |
| | 12.2 | Figures Shells | 39 |
| | | Section 14 Summary Tables Shells | |
| 13 | LIST | ING SHELLS | 66 |

## 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the analysis and presentation of the data from this study. Any changes made from the planned analysis described in the protocol or after finalization of this SAP will be documented in the Clinical Study Report (CSR). The section referred to as "Table, Figure, and Listing Shells" within this SAP describes the Clinical Data Interchange Standards Consortium (CDISC) input in order to provide traceability to the corresponding tables, figures, and listings (TFLs). Analysis data model (ADaM) is the source for tables and figures (as well as listings that may contain derived data) and study data tabulation model (SDTM) is the source for the data listings.

Any additional exploratory analyses not addressed within this SAP and/or driven by the data, or requested by the Philip Morris Products S.A., will be considered out of scope and must be described in the CSR.

#### 2. OBJECTIVES AND ENDPOINTS

| Endpoints |
|---|
| na nicotine concentration-time PK neters (THS regular stick, THS hol stick, and CIG separately): ximum nicotine plasma entration [Cmax] ne to the maximum nicotine plasma entration [Tmax] a under the curve of nicotine plasma entration-time computed from T0 to hours [AUC0-24h] a under the curve of nicotine plasma entration-time computed from T0 to ubject-specific time of maximum ine concentration [AUC0-Tmax] |
| nichine aa |

THS Induction device and regular or menthol sticks, P1-PK-12

# CA39924

| Secondary | |
|---|---|
| To evaluate pharmacodynamic (PD) effects (subjective effects) of a single use of a THS with either a regular or a menthol stick or of a single CIG. | <ul> <li>Score of CIG craving by the visual analogue scale (VAS) Craving assessment</li> <li>Score of investigational product (IP) liking by the VAS Liking assessment</li> <li>Score of intention to use the IP again by the VAS Intention to Use Again assessment</li> </ul> |
| To evaluate the safety of test products during the study. | <ul> <li>Incidence of adverse events (AEs) and serious adverse events (SAEs)</li> <li>Incidence of product events</li> <li>Changes in electrocardiogram (ECG) from baseline (heart rate, PR, QRS, QT, QTcF interval)</li> <li>Changes in vital signs from baseline (systolic and diastolic blood pressure, pulse rate and respiratory rate)</li> <li>Concomitant medication</li> <li>Changes in standard spirometry from baseline (FEV1, FEV1 % predicted, FVC, FVC % predicted, FEV1/FVC)</li> <li>Changes from baseline in clinical chemistry, hematology, and urine analysis safety panel</li> </ul> |

## 3. STUDY DESIGN

This study is designed to meet the objectives outlined in Section 2.

This is a single-center, randomized, controlled, open-label, cross-over study in healthy subjects. The study will be conducted with 3 periods and 6 sequences in a cross-over design.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

**Figure 1 Study Design** 



Abbreviations: CIG = combustible cigarette; P1M = menthol taste; P1R = regular taste

A Screening visit will be conducted within 27 days (Day -28 to Day -2) prior to admission (on Baseline Day -1) to the investigational site (Figure 1) to check and document the eligibility of the subjects. Investigational site staff will demonstrate the THS (without product use) during the Screening visit. The brand of subjects' cigarettes will be recorded.

Qualified subjects will return to the investigational site for Baseline on Day -1. Subjects will have fasted for at least 6 hours prior to the safety laboratory assessments. After confirmation of eligibility, subjects can be randomized. All subjects who will not be randomized will be documented as screen failures.

Thirty subjects will be randomized to one of 6 possible full crossover sequences of IP use (THS with either regular or menthol stick, and CIG) on Day 1 to Day 3 (see Figure 1). After admission on Baseline Day -1 in the morning, nicotine wash-out will start, and the use of any other tobacco and/or nicotine containing products (TNP) different from the IP assigned for use on Day 1 to Day 3, will not be allowed. Use of TNP will not be restricted after the subject has been discharged from the investigational site on Day 3.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

On Day 1 to Day 3, after at least 23 hours of abstinence from any TNP on Day 1, and after at least 24 hours of former IP use on Day 2 and Day 3 (nicotine wash-out), subjects will smoke a single CIG or perform a single use of a THS either with a regular or a menthol stick, according to randomized product use sequence.

The start of IP use will be defined as T<sub>0</sub>. T<sub>0</sub> on Day 1 to Day 3 should be at approximately the same time in the morning. Venous blood samples will be obtained according to the standard operating procedures (SOPs) at the investigational site. Subjects will report their cigarette craving, IP liking, and intention to use again by performing VAS assessments.

After Discharge on Day 3 or after Early termination following product exposure, the subjects will enter a 3-day Safety follow-up (SFU) period during which AE/SAEs reported by the subjects will be collected and the follow-up of AEs/SAEs will be conducted, concluded per a telephone contact by the investigational site on the last day of the SFU period.

#### 4. ANALYSIS POPULATIONS

## 4.1 Screened Population

The screened population consists of all subjects who underwent at least one screening procedure.

# 4.2 Safety Population (SAF)

The safety population is a subset of the screened population and consists of all subjects who give informed consent and have at least one safety assessment.

#### 4.3 Randomized Population

The randomized population is a subset of the safety population and consists of all the subjects who were randomized at Baseline (Day -1). Subjects for which inclusion/exclusion criteria were violated or subject for which the documentation for eligibility was incomplete at time of enrolment will be excluded from this population.

#### 4.4 Pharmacokinetic Population

The PK population is a subset of the randomized population and consists of all randomized subjects for whom at least one nicotine PK parameter can be derived. This population will also be applied for the PD parameters. Only subjects without major protocol deviations (see Section 4.4.1) which have an impact on evaluability of the main objective will be included in the PK population.

#### 4.4.1 Protocol Deviations

Protocol deviations are considered as deviations from the study procedures as defined in the study protocol, including but not limited to, as any violation of inclusion/exclusion criteria, mis-randomizations, assessments not performed or performed outside the scheduled time

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

windows, or use of drugs that are known to affect components of the "smokers' health profile."

Major protocol deviations are a subset of protocol deviations that may significantly impact the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being.

Subjects with major protocol deviations will be identified to determine whether they will be excluded from any of the analysis populations.

Major deviations will include but are not limited to the deviations presented in Table 4.1.

**Table 4.1 Definition of Major Protocol Deviations Categories** 

| Sub-Category | Description |
|---|---|
| Protocol violation | Violation of inclusion/exclusion criteria. Or missing documentation of any of the inclusion/exclusion criteria at time of enrollment. |
| Procedural deviation | Deviation to any study procedures. |
| Mis-randomization | Misclassification of subject's sex at randomization. Or incorrect product administered according to randomized sequence. |
| Use of TNP not allowed | Use of any nicotine or tobacco–containing product other than the assigned product during the exposure period, or use of any nicotine tobacco-containing product during at least 23 hours of abstinence from any nicotine/tobacco containing products (nicotine wash-out). |

#### 5. PRODUCT DESCRIPTIONS

#### 5.1 Test Products

Test product will be the THS induction device with regular and menthol sticks, provided by the Sponsor. The following two stick variants will be investigated:

| Name in the study (sticks) | Flavor |
|----------------------------|---------|
| P1R stick | Regular |
| P1M stick | Menthol |

The test products will be listed as:

| Name in the study (test products) | Abbreviated name (test products) |
|-----------------------------------|----------------------------------|
| THS regular stick (P1R) | P1R |
| THS menthol stick (P1M) | P1M |

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

# **5.2** Comparator Product

The subjects will bring their own supply of commercially available single brand CIG for the study duration.

The comparator product will be listed as:

| Name in the study (comparator product) | Abbreviated name (comparator product) |
|---|---|
| Combustible cigarette | CIG |

All subjects eligible at Screening visit and invited for Baseline visit Day -1 will be asked to purchase their usual brand of CIG and to provide it to the site personnel at their admission on Baseline (Day -1). Every subject will bring an unopened pack of CIG which will be kept in secured storage room at site with access limited to authorized personnel.

#### 6. PHARMACOKINETIC ANALYSIS

#### 6.1 Collection Schedule for Plasma Nicotine

Collection schedule is described in Table 6.1.

**Table 6.1 Plasma Nicotine Samples Collection Schedule** 

| Day 1<br>(14 blood<br>samples) | Prior to the start of product use $(T_B0) \le 5 \min (\pm 2 \min)$ prior to T0. In relation to T0 from Day 1: $T_B1$ after 4 minute $\pm$ 30 seconds, $T_B2$ after 6 minutes $\pm$ 1 minute, $T_B3$ after 8 minutes $\pm$ 1 minute, $T_B4$ after 10 minutes $\pm$ 1 minute, $T_B5$ after 12 minutes $\pm$ 1 minute, $T_B6$ after 15 minutes $\pm$ 2 minutes, $T_B7$ after 30 minutes $\pm$ 5 minutes, $T_B8$ after 1 hour $\pm$ 5 minutes, $T_B9$ after 2 hours $\pm$ 5 minutes, $T_B10$ after 4 hours $\pm$ 5 minutes, $T_B11$ after 10 hours $\pm$ 5 minutes, $T_B12$ after 14 hours $\pm$ 5 minutes, $T_B13$ after 24 hours $\pm$ 10 minutes |
|---|---|
| Day 2 | Same time points from T <sub>B</sub> 1 to T <sub>B</sub> 13. |
| (13 blood | T <sub>B</sub> 0 for Day 2 will be the same sample taken as T <sub>B</sub> 13 on Day 1. |
| samples) | |
| Day 3 | Same time points from T <sub>B</sub> 1 to T <sub>B</sub> 11 and no samples for T <sub>B</sub> 12, T <sub>B</sub> 13. |
| (11 blood | T <sub>B</sub> 0 for Day 3 will be the same sample taken as T <sub>B</sub> 13 on Day 2. |
| samples) | |

#### **6.2** Plasma Nicotine Concentrations

## Analytical Laboratory

Samples will be analyzed for nicotine in plasma using a validated liquid chromatography coupled to tandem mass spectrometry (LC-MS/MS) detection analytical method with the appropriate quality controls in accordance with the Food and Drug Administration (FDA)

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Guidance for Industry: Bioanalytical Method Validation (May, 2001) and in accordance with FDA Good Laboratory Practice regulations (Title 21 CFR Part 58) at Bioanalytical Services Lincoln, Nebraska.

#### 6.3 Plasma Nicotine Pharmacokinetic Parameters

Nicotine PK endpoints will be derived from measured plasma nicotine concentration-time data. Nicotine PK parameters will be derived using a non-compartmental analysis (NCA) technique using appropriate and validated PK software (e.g., Phoenix WinNonlin version 8.3.4 or higher).

For values above the upper limit of quantification (ULOQ), the ULOQ will be used for calculation and reporting in summary tables. For nicotine concentrations below the LLOQ (BLQ) for the calculation of descriptive statistics of observed plasma nicotine concentrations: In general, BLQ values before T0 will be imputed by LLOQ/2.

Plasma concentrations as determined at the collection times described in Section 6.1 will be used for the calculation of the plasma nicotine PK parameters.

BLQ values after the last quantifiable value are not included in the analysis (e.g., for the calculation of AUC).

Any BLQ value (after T0 and before the last quantifiable value) would need to be queried\* and, if confirmed, it will be imputed by LLOQ/2.

\*The query will be triggered at the latest by data QC, and will query the bioanalytical laboratory. The information on the value queried and a summarized response from the bioanalytical laboratory will be part of the SDTM data (e.g. in the CO domain).

The number and percent of values below LLOQ or above ULOQ will be presented in each summary table. If 50% or more data are below LLOQ or above ULOQ, only the number and percent of values below LLOQ or above ULOQ will be reported in the summaries, together with minimum (= LLOQ/2) and maximum (= ULOQ) of the observed values.

In particular, the following PK parameters will be derived from measured nicotine concentration-time data following IP use:

Cmax Maximum nicotine plasma concentration. Cmax will be reported as long

as there is at least one quantifiable concentration post T0.

Tmax Time to maximum nicotine plasma concentration Cmax.

AUC0-24 Area under the curve of nicotine plasma concentration-time computed

from T0 to T=24 hours [AUC0-24h].

AUC0-Tmax Area under the curve of nicotine plasma concentration-time computed

from T0 to the subject-specific time of maximum nicotine concentration

[AUC0-Tmax].

All AUC parameters will be calculated using linear trapezoidal with linear interpolation method.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

For PK analyses, baseline (pre-product use concentration) will be defined as the last assessment prior to T0 (5 minutes prior to T0) for each study day of exposure. PK parameters will not be calculated for subjects with less than 3 consecutive post-product use time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables and individual concentration-time figures only and excluded from the summary and statistical analysis.

#### 6.4 Data Summarization and Presentation

SAS software (version 9.4, Cary, North Carolina) will be used for all data presentation and summarization including statistical analyses, summary tables, graphs, and data listings.

All data will be presented in listings, ordered by subject, study visit, IP, and time point, unless otherwise specified.

PK data will be summarized for the PK population. In addition, PK data will also be summarized for the randomized population if there is at least a difference of 1 subject between the populations.

The 95% confidence interval (CI) of the arithmetic mean, median, first and third quartiles, minimum, maximum; for log-normal data, the geometric mean, geometric coefficient of variation (CV), and 95% CI of the geometric mean will be presented instead of arithmetic mean, SD, and 95% CI of the arithmetic mean, respectively.

For log normally distributed endpoints (Cmax, AUC0-24h and AUC0-Tmax), geometric mean, geometric CV, and confidence interval will be presented additionally.

Measured plasma nicotine concentrations and derived PK parameters will be summarized with descriptive statistics including number of subjects (n), number and percent of subjects with missing data (Missing, n (%)), arithmetic mean (Mean), arithmetic standard deviation (SD), 95% confidence interval (95%CI), minimum, first quartile (Q1), median, third quartile (Q3), and maximum. Summaries will be further stratified by Sex.

For log normally distributed endpoints (Cmax, AUC0-24h and AUC0-Tmax), geometric mean (Geo. Mean), 95% geometric confidence interval (Geo. 95% CI) and geometric CV (Geo. CV%) will be presented additionally.

For observed plasma nicotine concentrations, the number and percent of values below LLOQ (BLQ, n(%)) or above ULOQ (ALQ, n(%)) will be presented in each summary table.

Ordinal categorical data (e.g., Tmax) will be summarized by number of subjects (n), number and percent of subjects with missing data, median, first and third quartiles, and minimum and maximum.

All PK analyses and summaries will be performed by product.

The analytical data will be presented in the tables/listings to the same precision as received from the analytical laboratory.

The level of precision will be presented as follows: minimum/maximum in the same precision as in the database, mean/median in one more precision level than minimum/maximum, SD in

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

one more precision level than mean/median, and n will be presented as an integer. Percentages will be presented as an integer.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators. Missing PK data will be treated as missing and no data imputation will be conducted.

Mean and individual plasma nicotine concentrations will be presented graphically (linear and semi-log plots; linear plots will be presented with and without SD).

# 6.5 Statistical Analysis of Pharmacokinetic Parameters

## 6.5.1 Main Analysis

A mixed model analysis of variance (ANOVA) will be conducted on Cmax, AUC0-24h, and AUC0-Tmax endpoints in the natural logarithmic scale.

The model will include terms for sequence, period, product as fixed effects and subject as a categorical random effect modeling the within subject correlations.

The ANOVA analysis could be performed using the following SAS code:

```
PROC MIXED data=<> method=REML; class subject sequence period product; model log(parameter) = sequence period product/ddfm=KR; repeated product / subject=subject type=csh; lsmeans product / pdiff=control("CIG") cl alpha=0.05; RUN:
```

The results of this analysis for each of are presented in terms of geometric least square ratios and 95% confidence intervals for each THS / CIG ratio.

This approach is consistent with the guidelines in the European Medicines Agency's guidelines for bioequivalence investigations and FDA's Center for Drug Evaluation and Research.

The analysis of Tmax will be performed by conducting a Wilcoxon signed rank test and calculating the median Tmax for each product along with the Hodges-Lehmann estimate of the median difference between products, and the related 95% CI.

This analysis could be performed using the following SAS code:

```
PROC NPAR1WAY hl(refclass=<>) alpha=.05 data=<> hl; class TRT; var AVAL; ods output HodgesLehmann=HodgesLehmann; RUN;
```

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

## 6.5.2 Sensitivity Analyses

In case of any uncorrected nicotine concentration at T<sub>0</sub> [uC<sub>0</sub>] greater than 5% of their uncorrected maximum value, a sensitivity analysis of the PK endpoints will be performed similarly to the main analysis, whereby data of these subjects for this specific study day will be excluded from the analysis.

# 6.5.3 Supplementary Analysis

No supplementary analysis is foreseen.

#### 6.6 Preliminary Data and Interim Analysis

Biometrics will not perform preliminary or interim analyses.

### 7. PHARMACODYNAMIC EFFECTS (SUBJECTIVE EFFECTS)

#### 7.1 Data Collection

On Day 1 to Day 3, cigarette craving, product liking, and intention to use the product again will be assessed using a VAS (a 100 mm unipolar scale going from "no craving" to "strong craving" for VAS Craving; a 100 mm bipolar scale going from "strong disliking" to "strong liking" for VAS Liking; and a 100 mm bipolar scale going from "very unlikely" to "very likely" for VAS Intention to Use Again) at the following time points in relation to T0 with a time window as indicated in brackets:

#### Prior to T0 (for VAS Craving assessment)

• Tv0: within 15 minutes prior to T0

#### After T0 (for VAS Craving assessment)

- Tv1 after 4 minutes (± 2 minutes)
- Tv2 after 10 minutes ( $\pm$  2 minutes)
- Tv3 after 15 minutes (± 2 minutes)
- Tv4 after 30 minutes (± 2 minutes)
- Tv5 after 10 hours (± 5 minutes)

#### After T0 (for VAS Liking and VAS Intention to Use Again assessments)

• Tv3 after 15 minutes (± 1 minute)

#### 7.2 Data Summarization

Descriptive statistics (n, mean, SD, CV%, SEM, minimum, Q1, median, Q3, maximum, and 95% CI of mean) for VAS Craving assessment, VAS Liking assessment, and VAS

Intention to Use Again assessment will be provided by IP and assessment time point, as applicable. Change from baseline (pre-product use) for VAS Craving score will be summarized by IP and assessment time point. Individual responses will be listed. Summaries will be further stratified by sex.

PD data will be summarized for the PK population. In addition, PD data will also be summarized for the randomized population if there is at least a difference of 1 subject between the populations.

#### 8. SAFETY

All relevant case report form (CRF) data will be listed by subject and chronologically by assessment time point. This will include rechecks, unscheduled, and early termination assessments.

Applicable continuous variables will be summarized using n, mean, SD, minimum, median, and maximum.

The level of precision will be presented as follows: minimum/maximum in the same precision as in the database, mean/median in one more precision level than minimum/maximum, SD in one more precision level than mean/median, and n will be presented as an integer. Percentages will be presented as an integer.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

Baseline will be the result closest and prior to the product use in the respective period unless otherwise stated. Summaries for post-baseline time points will not include rechecks, unscheduled, or early termination measurements.

Tables summarizing safety data by assessment time point will only include summaries for baseline and post-baseline time points.

# 8.1 Subject Disposition

Subjects will be summarized by number of subjects screened, enrolled, enrolled and exposed to P1 product, randomized, completed, and discontinued the study with discontinuation reasons.

#### **8.2** Protocol Deviations

Protocol deviations are captured by the clinical site and provided in the CSR in a similar format to that provided by the clinical site. Protocol deviations are not edited or processed in SAS®.

## 8.3 Demographics

Descriptive statistics will be calculated overall for continuous variables (age, weight, height, and body mass index) and further stratified by sex.

Frequency counts will be provided for categorical variables (race, ethnicity, and sex) overall and further stratified by sex.

Demographic information and baseline characteristics (weight, height, and body mass index [BMI]) will be summarized for the safety and PK population. This summary will also be performed for the randomized population if there is at least a difference of 1 subject between the populations.

## 8.4 Tobacco/Nicotine-Containing Product Use History Questionnaire

At the Screening Visit, subjects will be asked questions about their tobacco-and/or nicotine-containing product (TNP) use history. The questions will capture frequency and quantity of TNP use over the past 4 weeks, and number of continuous years of cigarette smoking.

Descriptive statistics will be calculated for continuous variables overall and further stratified by sex.

Frequency counts and percentage will be provided for categorical variables overall and further stratified by sex.

## 8.5 Usual Brand Cigarettes Documentation

Subject's usual brand of cigarettes will be documented and frequency counts will be provided for categorical variables (substance, brand, brand style, flavor, and cigarette length) overall and further stratified by sex. Descriptive statistics will be presented for amount of use overall and further stratified by sex.

## 8.6 Fagerström Test for Nicotine Dependence (FTND)

Potential nicotine dependence will be assessed at the Screening Visit using the FTND in its revised version as updated in 2012 (Fagerström, K.O., 1978, Heatherton, T.F., et al., 1991). The questionnaire consists of six questions, which have to be answered by the subject himself/herself. The total score obtained on the test permit the classification of nicotine dependence into three levels: Mild (0 to 3 points); Moderate (4 to 6 points); Severe (7-10 points) (Fagerström, K., et al., 2012).

Descriptive statistics will be calculated for FTND score. In addition, frequency counts will be provided for nicotine dependence levels (mild, moderate, and severe) overall and further stratified by sex.

# 8.7 Medical History

All Medical History and Concomitant Disease will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 25.1 and listed by subject.

#### 8.8 Adverse Events

All AEs occurring during this clinical trial will be coded using MedDRA®, Version 25.1.

All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, product, severity, relationship to study product, and action; however, only product use-emergent AEs (PUEAEs) will be summarized. Adverse events after ICF and prior to the first product use on Day 1 and occurred during SFU period (after discharge from CRU to SFU visit) will be summarized separately under admission/SFU period.

A PUEAE is defined as an AE that is starting or worsening at the time of or after first study product administration. An AE that occurs during the washout period between study products is considered study product use emergent to the last study product given.

If the onset time of an AE is missing and the onset date is the same as the product administration date, the AE will be considered product use-emergent to the prior and current product. If the onset time of an AE is missing and the onset date does not fall on a product administration date, the AE will be considered product use-emergent for the last product administered. If the onset date of an AE is missing, the AE will be considered product use-emergent and attributed to each product on the study, unless the onset date is known to have occurred within or between specific product periods.

The number and percentage of subjects with AEs, SAEs will be tabulated by system organ class and preferred term. Summaries will also be presented for AEs leading to discontinuation, AEs leading to death, AEs by relatedness to product exposure, AEs by severity, and laboratory AEs. Tabulations will be performed for both the number of subjects experiencing an event and the number of events.

SAEs, if present, will also be listed. Applicable narratives will be included in the CSR.

# 8.9 Clinical Laboratory Tests (Serum Chemistry, Hematology, and Urinalysis)

Clinical laboratory evaluations (clinical chemistry, hematology, and urinalysis) will be performed at Screening, Admission (Day -1), and at the time of discharge (Day 3) or as early termination assessments, as applicable.

Out-of-normal range flags will be recorded as follows: high (H) and low (L) for numerical results and did-not-match (\*) for categorical results. If a value fails the reference range, it will automatically be compared to a computer clinically significant (CS) range. If the value falls within the computer CS range, it will be noted as "N" for not clinically significant. If the value fails (i.e., fall outside of the CS range) the computer CS range, it will be flagged with a

"Y" which prompts the PI to determine how the out-of-range value should be followed using 4 Investigator flags: "N", not clinically significant, "R", requesting a recheck, "^", checking at the next scheduled visit, or "Y", clinically significant. To distinguish the PI flag from the computer CS range flags, the PI flags of "N" and "Y" will be presented as "-" and "+", respectively, in the data listing. Additionally, a derived flag based on a search of the PI comments for a comment of "CS" or "Clinically Significant" will be used. The derived flag will be populated with "+" if the positive clinically significant determination is found in the comments for cases when the PI flag is populated with a "^" or a "R".

Out-of-range values and corresponding recheck results will be listed. CTCAE laboratory grading (version 5.0) will be included as well. Other lab results within this panel and time point will also be listed for this subject. Results that are indicated as CS by the PI will be listed in the table.

For all numeric laboratory values, descriptive statistics will be presented for each laboratory test by time point (baseline and discharge). Change from baseline will be summarized in a similar manner. Baseline is defined as the result closest and prior to the first product administration, which may include unscheduled or recheck results. This will typically be the result collected on Admission (Day -1). Post product use unscheduled events or rechecks will not be included in summaries. Similarly, early termination results will not be included in summaries.

# 8.10 Vital Signs

Vital signs (systolic and diastolic blood pressure, pulse rate, and respiratory rate) will be measured at the Screening Visit, on Admission (Day -1), Preuse on Period 1, Period 2, and Period 3, and Discharge (Period 3) or as early termination assessments, as applicable. All parameters will be recorded in supine position after the subject has rested for at least 5 minutes. Subjects should have abstained from using any TNPs for at least 15 minutes prior to Vital signs assessment.

The Investigator will define vital sign ranges to determine normal or abnormal results. For those results outside of the normal range, the Investigator will determine appropriate follow up including reporting of any AEs.

Descriptive statistics will be reported for vital signs measurements (blood pressure, pulse, respiration, and temperature) by time point. Change from baseline will be summarized in a similar manner. Baseline is defined as the result closest and prior to the first product administration, which may include unscheduled or recheck results. This will typically be the result collected on prior to T0 on Day 1. Post product use unscheduled events or rechecks

will not be included in summaries. Similarly, early termination results will not be included in summaries.

#### 8.11 Electrocardiogram

An ECG will be recorded at Screening, Admission (Day -1), and at discharge or at early termination. The ECG testing will be performed as per the investigational site standard practice. A standard 12-lead ECG will be recorded after the subject has rested for at least 10 minutes in supine position.

The following parameters will be documented: heart rate, PR interval, QRS interval, QT interval, and QTc interval, corrected by the ECG device according to Fridericia's formula [QTcF]. Each ECG will be assessed as normal, abnormal – not clinically significant, or abnormal – clinically significant.

Descriptive statistics will be presented for each ECG parameter by time point. Change from baseline will be summarized in a similar manner. Baseline is defined as the result closest and prior to the first product administration, which may include unscheduled or recheck results. This will typically be the result collected at Admission (Day -1). Post product use unscheduled events or rechecks will not be included in summaries. Similarly, early termination results will not be included in summaries.

#### 8.12 Prior and Concomitant Medications and Concomitant Procedures

All prior and concomitant medications will be listed by subject and product using Anatomical Therapeutic and Chemical (ATC) codes (World Health Organization Drug Dictionary) Version 01 Sep 2022 b3. Prior and concomitant medications concomitant procedures recorded during the study will be listed by subject.

#### 8.13 Physical Examination

A physical examination will be conducted at the Screening Visit. All data found in the CRF will be listed. Physical examination will be assessed as normal, abnormal – clinically not significant, or abnormal – clinically significant.

# 8.14 Spirometry

Spirometry without bronchodilator will be performed at the Screening Visit, Day -1, and at Discharge or early termination in accordance with the 2019 guideline update of the American Thoracic Society (ATS)/European Respiratory Society (ERS) Joint Task Force on the standardization of spirometry (Graham, B.L., et al., 2019). Spirometry predicted values will be standardized to the National Health and Nutrition Examination Survey III predicted set.

Assessed parameters will include: FEV1, FEV1% predicted, FVC, FVC% predicted, and FEV1/FVC.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Every Spirometry assessment has to be classified as normal, abnormal – clinically not significant, or abnormal – clinically significant.

Descriptive statistics will be presented for each spirometry parameter by time point. Change from baseline will be summarized in a similar manner. Baseline is defined as the result closest and prior to the first product administration, which may include unscheduled or recheck results. This will typically be the result collected at Day -1. Post product use unscheduled events or rechecks will not be included in summaries. Similarly, early termination results will not be included in summaries.

#### 8.15 Product Events

All product events occurring during this clinical trial will be collected and listed by subject.

#### 9. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol.

#### 10. REFERENCES

Committee for Medicinal Products for Human Use (CHMP) and European Medicines Agency (EMA), *Guideline on the investigation of bioequivalence* (CPMP/EWP/QWP/1401/98 Rev.1/Corr). 2010.

Fagerström, K.O., 1978

Fagerström, K.O., Measuring degree of physical dependence to tobacco smoking with reference to individualization of treatment. Addict Behav, 1978. 3(3-4): p. 235-41.

Fagerström, K., et al., 2012

Fagerström, K., et al., The Fagerström Test for Nicotine Dependence as a predictor of smoking abstinence: a pooled analysis of varenicline clinical trial data. Nicotine and Tobacco Research, 2012. 14(12): p. 1467-73.

FDA (Food and Drug Administration), *Guidance for industry – Statistical approaches to establishing bioequivalence.* 2001. Available from:

http://www.fda.gov/downloads/Drugs/.../Guidances/ucm070244.pdf (Accessed on 24 April 2014)

Heatherton, T.F., et al., 1991

Heatherton, T.F., et al., The Fagerström test for Nicotine Dependence: a revision of the Fagerström Tolerance Questionnaire. Br J Addict, 1991. 86(9): p. 1119-27.

Graham, B.L. et. al. 2019

Graham, B.L. et. al., Standardization of Spirometry 2019 Update. Am J Respir Crit Care Med Vol 200, Iss 8, pp e70–e88, Oct 15, 2019.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

### 11. SUMMARY TABLES, FIGURES, AND LISTINGS

Summary tables and figures are numbered following the International Council on Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using SAS® Version 9.4 or higher, as appropriate.

In-text tables and figures will be generated as RTF and all other tables and listings will be generated as SAS® LST format and converted to MS Word for inclusion in the CSR. In compliance SOP/PG, SAS® outputs will not be manually edited.

## 11.1 In-text Summary Tables and Figures

The following is a list of table and figure titles that will be included in the text of the CSR. Tables and figures will be numbered appropriately during compilation of the CSR.

#### Section 10:

| Number | Title | Shell |
|------------|-----------------------------------------|-------|
| Table 10-1 | Disposition Summary (Safety Population) | IDS |

#### **Section 11:**

| Number | Title | Shell |
|---|---|---|
| Table 11-1 | Summary of Demographics and Baseline<br>Characteristics (Safety Population) | IDEM |
| Table 11-2 | Summary of Plasma Nicotine PK Parameters of THS and CIG (PK Population) | ITPPar1 |
| Table 11-3 | Statistical Comparisons of Plasma Nicotine PK<br>Parameters for THS and CIG (PK Population) | ITPStat1 |
| Table 11-4 | Statistical Comparisons of Plasma Nicotine PK<br>Parameter Tmax for THS and CIG (PK Population) | ITPStat2 |
| Table 11-5 | Summary of VAS Craving Assessment (PK Population) | ITPDSum1 |
| Table 11-6 | Summary of VAS Liking Assessment (PK Population) | ITPDSum2 |
| Table 11-7 | Summary of VAS Intention to Use Again Assessment (PK Population) | ITPDSum2 |
| Figure 11-1 | Arithmetic Mean Plasma Nicotine Concentration<br>Versus Time Profiles Following Administration of<br>THS and CIG (Linear Scale) (PK Population) | PFPConc2 |

THS Induction device and regular or menthol sticks, P1-PK-12



## **Section 12:**

| Number | Title | Shell |
|---|---|---|
| Table 12-1 | Overall Product Use Emergent Adverse Events (Safety Population) | IAEO |
| Table 12-2 | Summary of Adverse Events by System Organ Class and Preferred Term (Safety Population) | IAES |

# 11.2 Section 14 Summary Tables and Figures

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be renumbered as appropriate during the compilation of the report.

## 14.1 Demographic Data Summary Tables

Note: Demographic TFLs may also include PK population. If so, the applicable titles will read: "Safety and PK Populations".

| Number | Title | Shell |
|---|---|---|
| Table 14.1.1 | Disposition Summary (Safety Population) | CDS |
| Table 14.1.2 | Subject Product Use Status and Study Disposition (Safety Population) | SDS |
| Table 14.1.3 | Demographic Summary (Safety Population) | CDEM |
| Table 14.1.4 | Tobacco/Nicotine-Containing Product Use History<br>Summary (Safety Population) | CUB |
| Table 14.1.5 | Usual Brand Cigarettes Summary (Safety Population) | CSU |
| Table 14.1.6 | Fagerstrom Test for Nicotine Dependence Summary (Safety Population) | CFT |

# 14.2 Pharmacokinetic/Pharmacodynamic Data Summary Tables and Figures

Note: PK and PD TFLs may also include Randomized population. If so, the applicable titles will read: "PK and Randomized Populations".

#### 14.2.1 Plasma Nicotine Tables

| Number | Title | Shell |
|---|---|---|
| Table 14.2.1.1 | Plasma Nicotine Concentrations (ng/mL) Following THS Regular stick (P1R) (PK Population) | CPCONC1 |

# THS Induction device and regular or menthol sticks, P1-PK-12

# CA39924

| Number | Title | Shell |
|---|---|---|
| Table 14.2.1.2 | Plasma Nicotine Concentrations (ng/mL) Following THS<br>Menthol stick (P1M) (PK Population) | CPCONC1 |
| Table 14.2.1.3 | Plasma Nicotine Concentrations (ng/mL) Following<br>Combustible Cigarette (CIG) (PK Population) | CPCONC1 |
| Table 14.2.1.4 | Plasma Nicotine Pharmacokinetic Parameters Following THS Regular stick (P1R) (PK Population) | CPPAR1 |
| Table 14.2.1.5 | Plasma Nicotine Pharmacokinetic Parameters Following THS Menthol stick (P1M) (PK Population) | CPPAR1 |
| Table 14.2.1.6 | Plasma Nicotine Pharmacokinetic Parameters Following<br>Combustible Cigarette (CIG) (PK Population) | CPPAR1 |
| Table 14.2.1.7 | Statistical Comparison of Plasma Nicotine<br>Pharmacokinetic Parameters: THS Versus CIG (PK<br>Population) | CPStat1 |
| Table 14.2.1.8 | Nonparametric Statistical Comparison of Plasma Nicotine<br>Tmax: THS Versus CIG (PK Population) | CPStat1 |

# 14.2.2 Plasma Nicotine Figures

| Number | Title | Shell |
|---|---|---|
| Figure 14.2.2.1 | Arithmetic Mean (SD) Plasma Nicotine Concentration<br>Versus Time Profiles Following Administration of THS<br>and CIG (Linear Scale) (PK Population) | PFPConc1 |
| Figure 14.2.2.2 | Arithmetic Mean Plasma Nicotine Concentration Versus<br>Time Profiles Following Administration of THS and CIG<br>(Linear Scale) (PK Population) | PFPConc2 |
| Figure 14.2.2.3 | Arithmetic Mean Plasma Nicotine Concentration Versus<br>Time Profiles Following Administration of THS and CIG<br>(Semi-Log Scale) (PK Population) | PFPConc3 |

# 14.2.3 Subjective Effects and Related Behavioral Assessment Tables

| Number | Title | Shell |
|---|---|---|
| Table 14.2.3.1 | Summary of VAS Craving Assessment by Study Product and Time Point (PK Population) | CPD1 |
| Table 14.2.3.2 | Summary of VAS Liking Assessment by Study Product (PK Population) | CPD1 |

# THS Induction device and regular or menthol sticks, P1-PK-12

# CA39924

| Number | Title | Shell |
|---|---|---|
| Table 14.2.3.3 | Summary of VAS Intent to Use Again Assessment by Study Product and Time Point (PK Population) | CPD1 |

# 14.3 Safety Data Summary Tables

# 14.3.1 Displays of Adverse Events

| Number | Title | Shell |
|---|---|---|
| Table 14.3.1.1 | Overall Product Use Emergent Adverse Event Frequency by Study Product – Number of Subjects Reporting the Event (% of Subjects Used IP) (Safety Population) | CAEO |
| Table 14.3.1.2 | Product Use Emergent Adverse Event Frequency by<br>Study Product – Number of Subjects Reporting the<br>Event (% of Subjects Used Study Product) (Safety<br>Population) | CAES |
| Table 14.3.1.3 | Product Use Emergent Serious Adverse Event Frequency by Study Product – Number of Subjects Reporting the Event (% of Subjects Used Study Product) (Safety Population) | CAES |
| Table 14.3.1.4 | Product Use Emergent Adverse Event Frequency by<br>Study Product – Number of Adverse Events (% of Total<br>Adverse Events) (Safety Population) | CAEE |
| Table 14.3.1.5 | Product Use Emergent Serious Adverse Event<br>Frequency by Study Product – Number of Adverse<br>Events (% of Total Adverse Events) (Safety Population) | CAEE |
| Table 14.3.1.6 | Product Use Emergent Adverse Event Frequency by<br>Study Product, Severity, and Relationship to Study<br>Product – Number of Adverse Events (Safety<br>Population) | CAESR |

# 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

| Number | Title | Shell |
|----------------|--------------------------------------------|--------|
| Table 14.3.2.1 | Serious Adverse Events (Safety Population) | 16.2.7 |

# 14.3.3 Narratives of Deaths, other Serious and Certain other Significant Adverse Events

# 14.3.4 Abnormal Laboratory Value Listing (each subject)

| Number | Title | Shell |
|---|---|---|
| Table 14.3.4.1 | Out-of-Range Values and Recheck Results – Serum Chemistry (Safety Population) | |
| Table 14.3.4.2 | Out-of-Range Values and Recheck Results – Hematology (Safety Population) | CLBO |
| Table 14.3.4.3 | Out-of-Range Values and Recheck Results – Urinalysis (Safety Population) | |
| Table 14.3.4.4 | Clinically Significant Values and Recheck Results (Safety Population) | CLBS |

# 14.3.5 Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

| Number | Title | Shell |
|---|---|---|
| Table 14.3.5.1 | Clinical Laboratory Summary and Change From Baseline – Serum Chemistry (Safety Population) | CLBD |
| Table 14.3.5.2 | Clinical Laboratory Shift From Baseline – Serum<br>Chemistry (Safety Population) | CLBS |
| Table 14.3.5.3 | Clinical Laboratory Summary and Change From Baseline – Hematology (Safety Population) | CLBD |
| Table 14.3.5.4 | Clinical Laboratory Shift From Baseline – Hematology (Safety Population) | CLBS |
| Table 14.3.5.5 | Clinical Laboratory Summary and Change From Baseline – Urinalysis (Safety Population) | CLBD |
| Table 14.3.5.6 | Clinical Laboratory Shift From Baseline – Urinalysis (Safety Population) | CLBS |
| Table 14.3.5.7 | Vital Sign Summary and Change From Baseline (Safety Population) | CVS |
| Table 14.3.5.8 | 12-Lead Electrocardiogram Summary and Change From Baseline (Safety Population) | CEG |
| Table 14.3.5.9 | Spirometry Summary and Change From Baseline (Safety Population) | CSP |

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

## 11.3 Section 16 Data Listings

Note: Hepatitis and HIV results that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in any database transfer. All data will be presented as outline in the CRF (i.e., time point information will be consistent with the CRF data).

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the TFLs for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

## **16.1** Study Information

#### 16.1.9 Statistical Methods

| Number | Title |
|-------------------|----------------------------------------|
| Appendix 16.1.9.1 | Statistical Analysis Plan |
| Appendix 16.1.9.2 | Statistical Methods – Pharmacokinetics |

### 16.1.10 Clinical Laboratory Reference Ranges

| Number | Title |
|--------------------|--------------------------------------|
| Appendix 16.1.10.1 | Clinical Laboratory Reference Ranges |

## 16.2 Subject Data Listings

#### **16.2.1 Subject Discontinuation**

| Number | Title |
|-------------------|-----------------------------------------|
| Appendix 16.2.1.1 | Subject Disposition (Safety Population) |
| Appendix 16.2.1.2 | Subject Disposition (Screen Failures) |

#### 16.2.2 Protocol Deviations

| Number | Title |
|-------------------|---------------------|
| Appendix 16.2.2.1 | Protocol Deviations |

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

# 16.2.3 Subjects Excluded From the Pharmacokinetic/Pharmacodynamic Analysis

| Number | Title |
|---|---|
| Appendix 16.2.3.1 | Subjects Excluded From the Pharmacokinetic/Pharmacodynamic Analysis |

Note: Appendices 16.2.2.1 and 16.2.3.1 are generated in MS Word for inclusion in the study report.

# 16.2.4 Demographic Data

| Number | Title |
|---|---|
| Appendix 16.2.4.1 | Demographics (Safety Population) |
| Appendix 16.2.4.2 | Demographics (Screen Failure) |
| Appendix 16.2.4.3 | Informed Consent (Safety Population) |
| Appendix 16.2.4.4 | Informed Consent (Screen Failure) |
| Appendix 16.2.4.5 | Physical Examination (I of II) (Safety Population) |
| Appendix 16.2.4.6 | Physical Examination (II of II) (Safety Population) |
| Appendix 16.2.4.7 | Physical Examination Descriptions (Safety Population) |
| Appendix 16.2.4.8 | Medical History (Safety Population) |
| Appendix 16.2.4.9 | Tobacco/Nicotine-Containing Product Use History (Safety Population) |
| Appendix 16.2.4.10 | Usual Brand Cigarettes Documentation (Safety Population) |
| Appendix 16.2.4.11 | Fagerstrom Test for Nicotine Dependence (Safety Population) |

## 16.2.5 Compliance and/or Concentration Data

| Number | Title |
|---|---|
| Appendix 16.2.5.1 | Subject Enrollment (Safety Population) |
| Appendix 16.2.5.2 | Subject Eligibility (Safety Population) |
| Appendix 16.2.5.3 | Subject Eligibility (Screen Failure) |
| Appendix 16.2.5.4 | Randomization (Safety Population) |
| Appendix 16.2.5.5 | Investigational Product Administration (Safety Population) |
| Appendix 16.2.5.6 | Prior and Concomitant Medications (Safety Population) |
| Appendix 16.2.5.7 | Plasma Nicotine Pharmacokinetic Blood Draw Times and<br>Concentration Data (Safety Population) |



# 16.2.6 Individual Pharmacokinetic/Pharmacodynamic Response Data

| Number | Title | Shell |
|---|---|---|
| Appendix 16.2.6.1 | Individual Plasma Nicotine Concentrations Versus Time for <subject #=""> (Linear and Semi-Log Scale)</subject> | PFPConc5 |
| Appendix 16.2.6.2 | VAS Craving Assessment (Safety Population) | |
| Appendix 16.2.6.3 | VAS Liking Assessment (Safety Population) | |
| Appendix 16.2.6.4 | Intention to Use Again (Safety Population) | |

## **16.2.7** Adverse Events Listings

| Number | Title |
|---|---|
| Appendix 16.2.7.1 | Adverse Events (Safety Population) |
| Appendix 16.2.7.2 | Details for Serious Adverse Events (Safety Population) This listing will be removed if no serious adverse events are reported. |
| Appendix 16.2.7.3 | Product Events (Safety Population) |

# 16.2.8 Clinical Laboratory Reports

| Number | Title |
|---|---|
| Appendix 16.2.8.1 | Clinical Laboratory Report - Serum Chemistry (Safety Population) |
| Appendix 16.2.8.2 | Clinical Laboratory Report - Hematology (Safety Population) |
| Appendix 16.2.8.3 | Clinical Laboratory Report - Urinalysis (Safety Population) |
| Appendix 16.2.8.4 | Clinical Laboratory Report - Urine Drug Screening (Safety Population) |
| Appendix 16.2.8.5 | Clinical Laboratory Report - Virology (Safety Population) |
| Appendix 16.2.8.6 | Alcohol Breath Test (Safety Population) |
| Appendix 16.2.8.7 | Vital Signs (Safety Population) |
| Appendix 16.2.8.8 | 12-Lead Electrocardiogram (Safety Population) |
| Appendix 16.2.8.9 | Spirometry (Safety Population) |

#### 12. TABLE, FIGURE, AND LISTING SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables that will be presented and included in the final report. Unless otherwise noted, all in-text tables will be presented in Times New Roman font size 9 and post-text tables will be presented in Courier New font size 9. In-text tables and figures will be generated as RTF and all other tables and listings will be generated as SAS® LST format and converted to MS Word for inclusion in the CSR. In compliance SOP/PG, SAS® outputs will not be manually edited.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

#### **In-text Summary Tables Shells** 12.1

In-text Shell IDS will be in the following RFT format:

# **Table IDS Disposition Summary (Safety Population)**

| Category | Overall |
|-------------------------------------|-----------|
| Screened | XXX |
| Enrolled | XX |
| Enrolled and Exposure to P1 Product | XX |
| Randomized | XX (100%) |
| Completed Study | XX (XX%) |
| Discontinued From Study | XX (XX%) |
| <reason></reason> | XX (XX%) |
| Source: Table 1/1 1 | |

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_disp.sas DDMMMYYYY HH:MM

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

In-text Shell IDM will be in the following RFT format:

**Table IDEM** Summary of Demographics and Baseline Characteristics (Safety Population)

| Trait | Category/Statistic | Overall |
|---------------|---------------------------|----------|
| Sex | Female | XX (XX%) |
| | Male | XX (XX%) |
| Race | Asian | XX (XX%) |
| | Black or African American | XX (XX%) |
| | White | XX (XX%) |
| Ethnicity | Hispanic or Latino | XX (XX%) |
| | Not Hispanic or Latino | XX (XX%) |
| Age (yr) | n | X |
| | Mean | X.X |
| | SD | X.XX |
| | Minimum | XX |
| | Median | X.X |
| | Maximum | XX |
| Body Mass | n | X |
| Index (kg/m²) | Mean | X.X |
| | SD | X.XX |
| | Minimum | XX |
| | Median | X.X |
| | Maximum | XX |
| Height (cm) | N | X |
| | Mean | X.X |
| | SD | X.XX |
| | Minimum | XX |
| | Median | X.X |
| | Maximum | XX |
| Weight (kg) | n | X |
| | Mean | X.X |
| | SD | X.XX |
| | Minimum | XX |
| | Median | X.X |
| | Maximum | XX |

Descriptive statistics for body mass index, height, and weight are calculated using Screening measurements.

Source: Table 14.1.3

Program: /CAXXXXX/sas prg/stsas/intext/t dem.sas DDMMMYYYY HH:MM

Programmer Note: If there is at least a difference of 1 subject between the safety, Randomized, and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.

In-text shell ITPPar1 will be in the following RFT format:

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

#### Table ITPPar1

## Summary of Plasma Nicotine PK Parameters of THS and CIG (PK Population)

| Pharmacokinetic Parameters | THS regular stick (P1R) | THS menthol stick (P1M) | Combustible Cigarette (CIG) |
|---|---|---|---|
| Param1 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param2 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param3 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param4 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |

Product <X>: <Label for Second Product>

Product <Y>: <Label for First Product >

Product <Z>: <Label for Third Product >

AUCs and Cmax values are presented as geometric mean and geometric CV%.

Tmax values are presented as median (min, max).

Source: Tables 14.2.1.4 through 14.2.1.6

#### Notes for Generating the Actual Table:

Presentation of Data:

- The following PK parameters will be presented in the following order and with following units: Cmax <ng/mL>, Tmax <min>, AUCO-24 <ng\*min/mL>, and AUCO-Tmax <ng\*min/mL>;
- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM

Programmer Note: If there is at least a difference of 1 subject between the Randomized and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

In-text shell ITPStat1 will be in the following RFT format:

#### **Table ITPStat1**

# Statistical Comparisons of Plasma Nicotine PK Parameters for THS and CIG (PK Population)

| | | | Product <y></y> | | | | |
|---|---|---|---|---|---|---|---|
| | Product <x> (Test)</x> | | (Comparator) | | | 95% Confidence | Intra subject |
| Parameter | Geometric LSMs | n | Geometric LSMs | n | GMR (%) | Interval | CV% |
| param1 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX | X.XX |
| param2 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX | X.XX |
| param3 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX | X.XX |

Product <X>: <Label for Test Product>

Product <Y>: <Label for Comparator Product >

Geometric least-squares means (LSMs) are calculated by exponentiating the LSMs derived from the ANOVA.

Geometric Mean Ratio (GMR) = 100\*(test/comparator)

Intra-subject CV% was calculated as 100 x square root(exp[MSE]-1), where MSE = Residual variance from ANOVA.

Source: Table 14.2.1.7

#### Notes for Generating the Actual Table:

Presentation of Data:

- The following PK parameters will be presented in the following order and with following units: Cmax (ng/mL), AUCO-24 <ng\*min/mL>, and AUCO-Tmax <ng\*min/mL>;
- n will be presented as an integer (with no decimal);
- All statistics will be presented with same precision as defined in post-text shells
- The comparisons will be: P1R vs CIG and P1M vs CIG, where P1R = THS regular stick; P1M = THS menthol stick; and CIG = Combustible cigarette.
- $\bullet\ \ \ \ \mbox{Add}$  column identifying the comparisons.

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam intext\_pkparam.sas DDMMYYYY HH:MM

Programming notes: The following comparisons will be included in the table: P1R versus CIG and P1M versus CIG.

If there is at least a difference of 1 subject between the Randomized and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

In-text shell ITPStat2 will be in the following RFT format:

#### **Table ITPStat2**

# Statistical Comparisons of Plasma Nicotine Pharmacokinetic Parameter Tmax for THS and CIG (PK Population)

| | | Difference <x> - <y></y></x> | | |
|---|---|---|---|---|
| Comparison | Parameter | Median | 95% Confidence Interval | p-value |
| P1R vs CIG | Tmax | X.XX | X.XX-X.XX | X.XXXX |
| P1M vs CIG | Tmax | X.XX | X.XX-X.XX | X.XXXX |

P1R: <> P1M: <> CIG: <>

The difference between products (product effect) and the 95% confidence interval for the difference was calculated using Hodges-Lehmann estimator.

Source: Table 14.2.1.8

#### Notes for Generating the Actual Table:

Presentation of Data:

- Median difference will be presented to 2 decimals or 3 significant figures
- 95% CI will be presented to 4 decimals
- p-value will be presented to 4 decimals

Programming notes: The following comparisons will be included in the table: P1R versus CIG and P1M versus CIG.

If there is at least a difference of 1 subject between the Randomized and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.

In-text Shell ITPDSum1 will be in the following RFT format:

## **Table ITPDSum1 Summary of VAS Craving Assessment (PK Population)**

| Time Point | THS regular stick (P1R) | THS menthol stick (P1M) | Combustible Cigarette (CIG) |
|---|---|---|---|
| Tv0: Within 15 minutes prior to T0 | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Tv1 after 4 minutes | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Tv2 after 10 minutes | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Tv3 after 15 minutes | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Tv4 after 30 minutes | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Tv5 after 10 hours | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Values are presented as arithmetic mean (± SD). | | | |
| Source: Tables <xxxx> and <yyyy></yyyy></xxxx> | | | |

Programmer Note: If there is at least a difference of 1 subject between the Randomized and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.
In-text Shell ITPDSum2 will be in the following RFT format:

## **Table ITPDSum2 Summary of VAS Liking Assessment (PK Population)**

| Time Point THS regular stick (P1R) | | THS menthol stick (P1M) | Combustible cigarette (CIG) |
|---|---|---|---|
| Tv3 after 15 minutes | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Values are presented as arithmetic mean (± SD). | | | |
| Source: Tables <xxxx> and <yyyy></yyyy></xxxx> | | | |

Programmer Note: If there is at least a difference of 1 subject between the Randomized and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

In-text Shell IAEO will be in the following RFT format:

## **Table IAEO** Overall Product Use Emergent Adverse Events (Safety Population)

| | | | Product Administration | | | |
|---|---|---|---|---|---|---|
| Adverse Event | Admission (N=X) | P1R (N = X) | P1M<br>(N-X) | CIG<br>(N = X) | Overall (N = X) | $ \mathbf{SFU} \\ (\mathbf{N} = \mathbf{X}) $ |
| Number of Subjects With PUEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects With SAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects With IP Events | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects With AEs Leading to Discontinuation | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects With AEs Leading to Death | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects With AEs Related to IP | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |

P1R: THS regular stick P1M: THS menthol stick CIG: Combustible cigarette

Although a subject may have had 2 or more adverse events, the subject is counted only once within a category. The same subject may appear in different categories.

PUEAEs = Product use-emergent adverse events; SAEs = Serious adverse events; IP = Investigational product

Admission = after ICF and prior to the product test on Day 1

SFU = after discharge from CRU to safety follow-up visit

Source: Table 14.3.1.1

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_ae.sas DDMMMYYYY HH:MM

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

In-text Shell IAES will be in the following RFT format:

Table IAES Summary of Adverse Events by System Organ Class and Preferred Term (Safety Population)

| | Admission | P1R | P1M | CIG | Overall | SFU |
|---|---|---|---|---|---|---|
| Adverse Event | (N=X) | (N = X) | (N-X) | (N = X) | (N = X) | (N = X) |
| Number of Subjects With PUEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects Without | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| PUEAEs | | | | | | |
| Eye disorders | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Visual blurred | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Gastrointestinal disorders | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Dyspepsia | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Nausea | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Musculoskeletal and connective tissue | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| disorders | | | | | | |
| Back pain | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Muscle cramps | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Musculoskeletal pain | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Nervous system disorders | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Headache | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Reproductive system and breast | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| disorders | | | | | | |
| Vaginal discharge | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Respiratory, thoracic and mediastinal | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| disorders | | | | | | |
| Epistaxis | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Skin and subcutaneous tissue | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| disorders | | | | | | |
| Sweating increased | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| D1D: THC regular stiels | | | | | | |

P1R: THS regular stick P1M: THS menthol stick CIG: Combustible cigarette

Although a subject may have had 2 or more adverse events, the subject is counted only once within a category. The same subject may appear in different categories.

Adverse events are classified according to MedDRA Version 25.1.

PUEAEs = Product use-emergent adverse events

Admission = after ICF and prior to the product test on Day 1

SFU = after discharge from CRU to safety follow-up visit

Source: Table 14.3.1.2

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_ae.sas DDMMMYYYY HH:MM

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

## 12.2 Figures Shells

Figures PFPConc2 (both in-text and post-text) will be in the following RFT format: Figure Mean Plasma Nicotine Concentrations Versus Time (Linear Scale) (PK Population)



Programming note: the legend will present the 3 products 'Product X: Product Description'

The x-axis title will be: 'Time From Start of Product Use (min)'.

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Figure PFPConc1 will be in the following RFT format:

Figure Mean (SD) Plasma Nicotine Concentrations Versus Time (Linear Scale) (PK Population)



Treatments B and C are shifted to the right for ease of reading

Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM

Program: /CAXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

Programming note: the legend will present the 3 products 'Product X: Product Description'

The x-axis title will be: 'Time From Start of Product Use (min)'.

CA39924

Figure PFPConc3 will be in the following RFT format:

Figure Mean Plasma Nicotine Concentrations Versus Time (Semi-Log Scale) (PK Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

Programming note: the legend will present the 3 products 'Time From Start of Product Use (min)'

The x-axis title will be: 'Time From Start of Product Use (min)'

# Linear and Semi-log Figures in Appendix 16.2.6.1 will have the following format:

Appendix 16.2.6.1

Individual Plasma Nicotine Concentrations Versus Time (Linear and Semi-Log Scales)



Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMMYYY HH:MM Programming note : the legend will present the 3 products. The x-axis title will be: 'Time From Start of Product Use (min)' The y-axis title will be: 'Plasma Nicotine Concentration (ng/mL)'

THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

# 12.3 Section 14 Summary Tables Shells

Table CDS Disposition Summary (Safety Population)

| Category | Overall |
|-------------------------------------|-----------|
| Screened | XXX |
| Enrolled | XX |
| Enrolled and Exposure to P1 Product | XX |
| Randomized | XX (100%) |
| Completed Study | XX (XX%) |
| Discontinued From Study | X ( XX%) |
| <reason></reason> | X ( XX%) |

Program: /CAXXXXX/sas\_prg/stsas/tab/programname2022Q1programname2022Q1.sas DDMMYYYY HH:MM


Table SDS Subject Product Use Status and Study Disposition (Safety Population) (Safety Population)

| 0.1.1 | | Randomized | Product Administrated | | inistrated | Study Completion | |
|---|---|---|---|---|---|---|---|
| Subject<br>Number | Product<br>Sequence | P1R | P1M | CIG | Status | Date | |
| | X | XXXXXXXXXX | Yes | No | Yes | Discontinued From Study: <reason></reason> | DDMONYYYY |
| | X | XXXXXXXXX | Yes | Yes | Yes | Completed Study | DDMONYYYY |
| | X | XXXXXXXXX | Yes | Yes | Yes | Completed Study | DDMONYYYY |
| | X | XXXXXXXXX | Yes | Yes | Yes | Completed Study | DDMONYYYY |
| | | | XX | XX | XX | | |

Programmer Note: Please refer to Section 5 for the product description.

P1R: < >

P1M: < > CIG: < >

 $\label{program: program: pro$ 

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Table CDEM Demographic Summary (Safety Population)


| Sex | Trait | Category/Statistic | Overall |
|---|---|---|---|
| All | Sex | Male<br>Female | X (XX%)<br>X (XX%) |
| | Race | Asian<br>Black or African American<br>White | X (XX%)<br>X (XX%)<br>X (XX%) |
| | Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | X (XX%) |
| | Age (yr) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X<br>X.X<br>X.XX<br>XX<br>XX<br>XX |
| | Body Mass Index (kg/m²) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | X X X X X X X X X X X X X X X X X X X |

Descriptive statistics for body mass index, height, and weight are calculated using screening measurements.

Program: /CAXXXXX/sas prg/stsas/tab/programname2022Q1.sas DDMMYYYYY HH:MM

Programmer note: If there is at least a difference of 1 subject between the safety, Randomized, and PK, and populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis. The summarization for each sex will also be presented.


Table CUB Tobacco/Nicotine-Containing Product Use History Summary (Safety and PK Population)

| Sex | Question | Product | Answer | Overall |
|---|---|---|---|---|
| All | Have you smoked continuously for the past 3 years? | Manufactured or roll-your-own cigarettes | Yes<br>No | X (XX.X%)<br>X (XX.X%) |
| | | Cigars/cigarillos | Yes<br>No | X(XX.X%)<br>X(XX.X%) |
| | xxxxx | XX | | |
| | In the last 4 weeks, on average how many of these products did you smoke/use per day? | Manufactured or roll-your-own cigarettes | 1 cigarette or less<br>2 to 5 cigarettes<br>6 to 9 cigarettes<br>10 to 19 cigarettes<br>1 to 2 packs<br>More than 2 packs | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%)<br>X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) |
| | Do you plan to quit smoking cigarettes within the next 3 months? | | Yes<br>No | X (XX.X%)<br>X (XX.X%) |
| | Do you plan to stop using tobacco and/or nicot containing products within the next 3 months? | | Yes<br>No | X(XX.X%)<br>X(XX.X) |

Program: /CAXXXXX/sas prg/stsas//tab/ADaM program name.sas DDMMMYYYY HH:MM

Programmer Note: All products (Manufactured or roll-your-own cigarettes, Cigars/cigarillos, Tobacco Pipe, Smokeless tobacco products, E-vapour products), and Nicotine replacement therapy (NRT) products in the tobacco/nicotine use history will be included in the descriptive statistics table. Number of years smoked will be presented using descriptive statistics. If there is at least a difference of 1 subject between the safety, Randomized, and PK, and populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis. The summarization for each sex will also be presented.


Table CSU Usual Brand Cigarettes Summary (Safety and PK Population)

| Sex | Trait | Category/Statistic | Overall |
|-----|------------------|-----------------------------------------|---------|
| All | Substance | XXXXX | X (XX%) |
| | | XXXXXXXXXX | X (XX%) |
| | Amount | n | X |
| | | Mean | X.X |
| | | SD | X.XX |
| | | Minimum | XX |
| | | Median | X.X |
| | | Maximum | XX |
| | Brand | XXXXXXXXX | X (XX%) |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X (XX%) |
| | | XXXXX | X (XX%) |
| | Brand Style | XXXXXXX | X (XX%) |
| | - | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X (XX%) |
| | Flavour | XXXXXXXXX | X (XX%) |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | Cigarette Length | XXXXXXXX | X (XX%) |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | X (XX%) |

Program: /CAXXXX/sas prg/stsas/tab/programname2022Q1.sas DDMMYYYY HH:MM

Programmer note: If there is at least a difference of 1 subject between the safety, Randomized, and PK, and populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis. The summarization for each sex will also be presented.

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Table CFT Fagerström Test for Nicotine Dependence Summary (Safety and PK Population)


| Sex | Trait | Category/Statistic | Overall |
|-----|---------------------------|--------------------|---------|
| All | Fagerstrom Score | n | X |
| - | - | Mean | X.X |
| | SD | | X.XX |
| | | Minimum | XX |
| | | Median | X.X |
| | | Maximum | XX |
| | Nicotine Dependence Level | Mild (0-3) | X (XX%) |
| | - | Moderate (4-6) | X (XX%) |
| | | Severe (7-10) | X (XX%) |

Program: /CAXXXXX/ sas prg/stsas/tab/programname2022Q1.sas DDMMYYYY HH:MM

Programmer note: If there is at least a difference of 1 subject between the safety, Randomized, and PK, and populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis. The summarization for each sex will also be presented.

## THS Induction device and regular or menthol sticks, P1-PK-12

### CA39924

### Note: Plasma Nicotine Concentration Tables (CPCONC1) will have the following format:


Table Plasma Nicotine Concentrations (ng/mL) Following THS Regular stick (P1R) (PK Population)

| Subject Product<br>Number Sequence | Sex | Pre-use | XX | XX | XX | Sample T<br>XX | imes (mir<br>XX | nutes)<br>XX | XX | XX | XX | XX |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XX XXXXXX<br>XX XXXXXX<br>XX XXXXXX | X<br>X<br>X | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX | XX<br>XX<br>XX |
| n n missing % n missing Mean SD 95% CI Minimum 1st quartile Median 3rd quartile Maximum | x. | X<br>X<br>X<br>X.X<br>X.X<br>X-X,X<br>X-X,X<br>XX<br>X.X<br>X.X<br>X.X | X<br>X<br>X.X<br>X.XX<br>X.X-X,X X<br>XX<br>X.X<br>X.X<br>X.X<br>X.X<br>X.X | X<br>X<br>X.X<br>X.XX<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X | X<br>X<br>X<br>X.X<br>X.X<br>X.X<br>XX<br>X.X<br>X.X<br>X.X<br>X.X | X<br>X<br>X.X<br>X.XX<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X<br>X.X | X<br>X<br>X.X<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X | X<br>X<br>X.X<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X | X<br>X.X<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X | X<br>X<br>X.X<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X | X<br>X.X<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X | X<br>X<br>X<br>X.X<br>X.XX<br>X.X-X,X<br>XX<br>X.X<br>X.X<br>X.X<br>X.X |

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming Notes: For the 95% CI (of Mean), the lower and upper limits may be presented on different rows if the space limit requires it. If there is at least a difference of 1 subject between the Randomized and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.

The number and percent of values below LLOQ or above ULOQ are to be presented in each summary table. If 50% or more data are below LLOQ or above ULOQ, only the number and percent of values below LLOQ or above ULOQ is to be reported in the summaries, together with minimum (= LLOQ/2) and maximum (= ULOQ) of the observed values.

Footnotes to include under the table, as appropriate:

<. = Concentration value missing or not reportable.>

<Concentration values that were below the limit of quantitation (BLQ) of 0.200 ng/mL were set to one-half of the limit of quantitation
for the calculation of summary statistics.>

Sample Times are listed in Section 6.1. Descriptive statistics precision is specified in Section 6.4.

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

### Note: Plasma Nicotine Pharmacokinetic Parameter Tables (CPPAR1) will have the following format:


Table Plasma Nicotine Pharmacokinetic Parameters Following THS Regular stick (P1R) (PK Population)

| Subject Product Sex | | | | | |
|---|---|---|---|---|---|
| Number Sequence | <unit></unit> | | | | |
| XX XXXXXX X | X.XX | | | | |
| XX XXXXXX X | X.XX | X.XX | X.XX | X.XX | X.XX |
| XX XXXXXX X | X.XX | X.XX | X.XX | X.XX | X.XX |
| n | X | X | Х | X | X |
| n missing | X | X | X | X | X |
| % n missing | X | X | X | X | X |
| Mean | X.X | X.X | X.X | X.X | X.X |
| SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| 95% CI of Mean | X.XX-XX.XX | (repeat | format | for other | parameters) |
| Minimum | XX | XX | XX | XX | XX |
| 1st quartile | X.X | X.X | X.X | X.X | X.X |
| Median | X.X | X.X | X.X | X.X | X.X |
| 3rd quartile | X.X | X.X | X.X | X.X | X.X |
| Maximum | XX | XX | XX | XX | XX |
| Geom. Mean | X.X | X.X | X.X | X.X | X.X |
| Geom. CV% | XX.X | XX.X | XX.X | XX.X | XX.X |
| 95% CI of Geom. Mean | X.XX-XX.XX | (repeat | format | for other | parameters) |

Program: /CAXXXXX/sas prg/pksas/PROGRAMNAME.SAS DDMMYYYYY HH:MM

Programming Notes: Footnote to include under the table, as appropriate: <. = Parameter value missing or not reportable.>
If there is at least a difference of 1 subject between the Randomized and PK populations, a column for population will be added as the first column and the summary statistics will be presented for each population with table title updated to reflect the populations used in the analysis.

The plasma nicotine PK parameters are Cmax (ng/mL), Tmax (min), AUCO-24 (ng\*min/mL), AUCO-Tmax (ng\*min/mL). Geometric mean, geometric CV% and 95% CI of Geom. Mean will be calculated only for Cmax, AUCO-24, and AUCO-Tmax.

For Tmax, only median, Q1, Q3, minimum and maximum will be presented.

Descriptive statistics precision is specified in Section 6.3.

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

## Note: Statistical comparison of PK parameters (CPStat1) will have the following format:


Table Statistical Comparison of Plasma Nicotine Pharmacokinetic Parameters Cmax, AUC0-24, and AUC0-Tmax (PK Population)

| Comparison | Parameter | Geometric<br>LS Means -<br>Test (n) Compa | arator (n) | % Geometric<br>LS Mean Ratio<br>(Test/Comparator) | 90% Confidence<br>Interval | p-value |
|---|---|---|---|---|---|---|
| P1R vs CIG | Cmax<br>AUCO-24<br>AUCO-Tmax | x.xx (x) x. | .XX (X)<br>.XX (X)<br>XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |
| P1M vs CIG | Cmax<br>AUCO-24<br>AUCO-Tmax | x.xx (x) x. | .XX (X)<br>.XX (X)<br>XX (X) | XXX.XX<br>XXX.XX<br>XXX.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X.XXXX<br>X.XXXX<br>X.XXXX |

P1R = < >

P1M = < >

 $CIG = \langle \rangle$ 

The mixed model includes sequence, period, product as fixed effects and subject as a categorical random effect modeling the within subject correlations.

Parameters are ln-transformed prior to analysis

Geometric least-squares means (LS Means) are calculated by exponentiating the LS Means from the ANOVA.

% Geometric LS Mean Ratio = 100\* (Test/Comparator)

Test = The first product in the comparison

Comparator = The second product in the comparison n = Number of observation used in the analysis

Program: /CAXXXXX/sas prg/pksas PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programming note: Geometric LS Means to be presented to same precision as Mean in the PK parameter table. Geometric Mean Ratio and 90% confidence intervals will be presented to 2 decimal places; p-value will be presented to 4 decimals.

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

# Note: Statistical comparison of PK parameter Tmax (CPStat2) will have the following format:


Table Statistical Comparison of Plasma Nicotine Pharmacokinetic Parameter Tmax (PK Population)

| | | Difference <x> - <y></y></x> | |
|-----------|--------|------------------------------|---------|
| Parameter | Median | 90% Confidence Interval | p-value |
| Tmax | x.xx | -x.xxxx - x.xxxx | X.XXXX |

Product: <Label for First Product >
Product: <Label for Second Product>

### Notes for Generating the Actual Table:

Presentation of Data:

- Median difference will be presented to 2 decimals or 3 significant figures
- 90% CI will be presented to 4 decimals
- p-value will be presented to 4 decimals

Programmers Note:

The comparisons will be: P1R vs CIG and P1M vs CIG, where P1R = THS regular stick; P1M = THS menthol stick; and CIG = Combustible cigarette. Add column identifying the comparisons.

The difference between products (product effect) and the 95% confidence interval for the difference was calculated using Hodges-Lehmann estimator.

Program: DM PX:[HLXXXXX.PKSAS]XXXX.SAS DDMMMYYYY HH:MM

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

# Note: Summary table (CPD1) will have the following format:

Table CPD1 Summary of VAS Craving Assessment by Study Product and Time Point (PK Population)

| | | | | Product | t |
|---------------|--------|--------------|---------|---------|---------|
| Time Point | Sex | Statistic | P1R | P1M | CIG |
| XXXXXXXXXXXXX | Female | n | Х | X | Х |
| | | Mean | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX |
| | | 1st quartile | X.X | X.X | X.X |
| | | Median | X.X | X.X | X.X |
| | | 3rd quartile | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX |
| | | 95% CI | X.X-X.X | X.X-X.X | X.X-X.X |
| | Male | n | X | X | X |
| | | Mean | X.X | X.X | X.X |
| | | SD | X.XX | X.XX | X.XX |
| | | CV (%) | XX.X | XX.X | XX.X |
| | | SEM | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX |
| | | 1st quartile | X.X | X.X | X.X |
| | | Median | X.X | X.X | X.X |
| | | 3rd quartile | X.X | X.X | X.X |
| | | Maximum | XX | XX | XX |
| | | 95% CI | X.X-X.X | X.X-X.X | X.X-X.X |

\_\_\_\_\_\_

P1R: < > P1M: < > CIG: < >

Program: /CAXXXXX/sas\_prg/pksas/PROGRAMNAME.SAS DDMMMYYYY HH:MM

Programmer Note: All collection time points and overall (sex combined) for each timepoint will also be presented in the table.

# THS Induction device and regular or menthol sticks, P1-PK-12 CA39924

Table CAEO Overall Product Use Emergent Adverse Event Frequency by Study Product - Number of Subjects Reporting the Event
(% of Subjects Used Study Product) (Safety Population)

#### Product Administration

| Adverse Event | Admission $(N = X)$ | P1R (N = X) | P1M $(N = X)$ | CIG $(N = X)$ | Overall $(N = X)$ | SFU<br>(N = X) |
|---|---|---|---|---|---|---|
| Number of Subjects With PUEAEs | X ( X%) | X ( XX%) | X ( XX%) | X ( X%) | X ( XX%) | X ( XX%) |
| Number of Subjects With SAEs | X ( X%) | X ( XX%) | X ( XX%) | X ( X%) | X ( XX%) | X (XX%) |
| Number of Subjects With IP Events | X ( X%) | X ( XX%) | X ( XX%) | X ( X%) | X ( XX%) | X (XX%) |
| Number of Subjects With AEs Leading to Discontinuation | X ( X%) | X ( XX%) | X ( XX%) | X ( X%) | X ( XX%) | X ( XX%) |
| Number of Subjects With AEs Leading to Death | X ( X%) | X (XX%) | X ( XX%) | X ( X%) | X ( XX%) | X ( XX%) |
| Number of Subjects With AEs Related to IP | X ( X%) | X ( XX%) | X ( XX%) | X ( X%) | X ( XX%) | X ( XX%) |

P1R: < > P1M: < > CIG: < >

Although a subject may have had 2 or more adverse events, the subject is counted only once within a category. The same subject may appear in different categories.

PUEAEs = Product use-emergent adverse events; SAEs = Serious adverse events; IP = Investigational product Admission = after ICF and prior to the product test on Day 1

SFU = after discharge from CRU to safety follow-up visit

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Table CAES Product Use Emergent Adverse Event Frequency by Study Product - Number of Subjects Reporting the Event
(% of Subjects Used Study Product) (Safety Population)

#### Product Administration

| | | | | | | SFU (N = X) X ( XX%) XX ( XX%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) |
|---|---|---|---|---|---|---|
| Adverse Event | Admission $(N = X)$ | P1R<br>(N = X) | P1M<br>(N = X) | CIG<br>(N = X) | Overall (N = X) | |
| Number of Subjects With PUEAEs Number of Subjects Without PUEAEs | X ( X%)<br>XX ( XX%) | X ( XX%)<br>XX ( XX%) | X ( XX%) | X ( X%)<br>XX ( XX%) | X ( XX%)<br>XX ( XX%) | , , |
| Eye disorders | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Vision blurred | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Gastrointestinal disorders | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Dyspepsia | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Nausea | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Musculoskeletal and connective tissue disorders | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Back pain | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Muscle cramps | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Musculoskeletal pain | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Nervous system disorders | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Headache | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Reproductive system and breast disorders | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Vaginal discharge | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Respiratory, thoracic and mediastinal disorders | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Epistaxis | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |

P1R: < > P1M: < >

CIG: < >

Although a subject may have had 2 or more adverse events, the subject is counted only once within a category. The same subject may appear in different categories.

Adverse events are classified according to MedDRA Version 25.1.

PUEAEs = Product use-emergent adverse events

 ${\tt Admission = after\ ICF\ and\ prior\ to\ the\ product\ test\ on\ Day\ 1}$ 

SFU = after discharge from CRU to safety follow-up visit


Table CAEE Product Use Emergent Adverse Event Frequency by Study Product - Number of Adverse Events (% of Total Adverse Events) (Safety Population)

| | | Pı | roduct Admin | istration | | |
|---|---|---|---|---|---|---|
| Adverse Event | Admission (N = X) | P1R<br>(N = X) | P1M<br>(N = X) | CIG<br>(N = X) | Overall<br>(N = X) | SFU<br>(N = X) |
| Number of PUEAEs | X ( X%) | , , | | X ( X%) | | X ( XX%) |
| Eye disorders Vision blurred Gastrointestinal disorders Dyspepsia Nausea Musculoskeletal and connective tissue disorders Back pain Muscle cramps Musculoskeletal pain | X ( X%) | X ( X%) | | X ( X%) | | X ( X%) |
| Nervous system disorders Headache Reproductive system and breast disorders Vaginal discharge Respiratory, thoracic and mediastinal disorders Epistaxis | X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) | X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) |

P1R: < > P1M: < > CIG: < >

Adverse events are classified according to MedDRA Version 25.1.

PUEAEs = Product use-emergent adverse events

 $\begin{array}{l} {\tt Admission = after\ ICF\ and\ prior\ to\ the\ product\ test\ on\ Day\ 1} \\ {\tt SFU = after\ discharge\ from\ CRU\ to\ safety\ follow-up\ visit} \\ \end{array}$ 


Table CAESR Product Use Emergent Adverse Event Frequency by Study Product, Severity, and Relationship to Study Product - Number of Adverse Events (Safety Population)

| | | Number of<br>Subjects<br>With | Number<br>of | | Severity | | _ | roduct | Relationshi<br>Study Proce | dure |
|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event | Product | PUEAEs | PUEAEs | Mild | Moderate | Severe | Unrelated | l Related | | Related |
| Abdominal pain | XXX | X | Х | Х | X | X | X | X | Х | X |
| Constipation | XXX | X | X | X | X | X | X | X | X | X |
| Dry throat | XXX | X | X | X | X | X | X | X | X | X |
| Dysmenorrhoea | XXX | X | X | X | X | X | X | X | X | X |
| Dyspepsia | XXX | X | X | X | X | X | X | X | X | X |
| Headache | XXX | X | X | X | X | X | X | X | X | X |
| | XXX | X | X | X | X | X | X | X | X | X |
| Myalgia | XXX | X | X | X | X | X | X | X | X | X |
| Nasal congestion | n XXX | X | X | X | X | X | X | X | X | X |
| Skin laceration | XXX | X | X | Χ | X | Χ | X | Χ | X | X |
| Adn | nission | Х | Х | Х | Х | X | X | Х | X | X |
| | P1R | X | X | X | X | X | X | X | X | X |
| | P1M | X | X | X | X | X | X | X | X | X |
| | CIG | X | X | X | X | X | X | X | X | X |
| ( | verall | X | X | X | X | X | X | X | X | X |
| | FU | X | X | X | X | Χ | X | X | X | X |

P1R: < > P1M: < >

CIG: < >

Adverse events are classified according to MedDRA Version 25.1.

PUEAEs = Product use-emergent adverse events

 ${\tt Admission = after\ ICF\ and\ prior\ to\ the\ product\ test\ on\ Day\ 1}$ 

SFU = after discharge from CRU to safety follow-up visit

Overall = From the product use on Day 1 through the discharge from CRU.


Table 14.3.2.1 Serious Adverse Events (Safety Population)

\_\_\_\_\_

Will match format of Appendix 16.2.7

Or contain statement as follows:

"There were no events that met this criteria."


Table CLBO Out-of-Range Values and Recheck Results - <Clinical Laboratory Panel> (Safety Population)

| Subject<br>Number | | 4 | Day | Hour | Date | Time | Parameter1<br><range><br/>(Unit)</range> | Parameter2<br><range><br/>(Unit)</range> | Parameter3<br><range><br/>(Unit)</range> | Parameter4<br><range><br/>(Unit)</range> |
|---|---|---|---|---|---|---|---|---|---|---|
| Χ Χ | XX/X | Screen<br>1 | -X | -x.xx | DDMMMYYYY<br>DDMMMYYYY | | XX HN<br>XX LN | XX LY- | XX LN G | 1 XX HN<br>XX LN |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early termination chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Unscheduled and Early Termination records should only be included if they are out of range or recheck results.

F = Female; M = Male H = Above reference range; L = Below reference rangeCS Flag: N = Not clinically significant; Y = Clinically significant PI interpretation: - = Not clinically significant CTCAE grade (Version 5.0): G1 = Mild

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Table CLBS Clinically Significant Laboratory and Corresponding Results (Safety Population)


| Subject Age/<br>Number Sex | - | Day Hour | Date | Time | Department | Test | Result | Reference Range | Unit |
|---|---|---|---|---|---|---|---|---|---|
| X XX/X | <br>: 1 | X -X.X D | DMMYYYY | HH:MM | Serum Chemistry | Cholesterol | XXX | x - x | mg/dL |

Programmer Note: All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table.

H = Above reference range

Computer: Y = Clinically significant

PI Interpretation: R = Recheck requested, + = Clinically significant

If no event meet this criteria then include a statement as follows:

"There were no clinical laboratory results documented as clinically significant by the PI."

# THS Induction device and regular or menthol sticks, P1-PK-12 CA39924

Table CLBD Clinical Laboratory Summary and Change From Baseline - <Clinical Laboratory Panel> (Safety Population)

Randomized Product Sequence XXX XXX Reference XXX XXX XXX XXX Laboratory Test (units) Range Time Point Statistic (N = X)(N = X)(N = X)(N = X)(N = X)(N = X)< - ># Χ Χ Χ Χ Χ Χ Testname (unit) Baseline n Mean X.X\* X.X X.X X.X X.X X.X\* SD X.XX X.XX X.XX X.XX X.XX X.XX Minimum XX XX XX XX XX XX Median X.X X.X X.X X.X X.X X.X Maximum XX XX XX XX XX XX Χ Χ Χ Χ Discharge Absolute Χ Χ X.X^ X.X X.X X.X^ X.X X.X Mean SD XX.XX XX.XX XX.XX X.XX X.XX X.XX Minimum XX XX XX XX XX XX Median X.X X.X X.X X.X X.X X.X Maximum XX XX XX XX XX XX Χ Χ Χ Χ Χ Change Χ Mean X.X^ X.X X.X X.X^ X.X X.X X.XX X.XX XX.XX X.XX X.XX X.XX SD Minimum XX XX XX XX XX XX Median X.X X.X X.X X.X X.X X.X

Programmer Note: Means at specific time points will be flagged (with a \*) if they are above or below the reference range. This only applies to the clinical laboratory results (i.e., not the change from baseline or any other endpoints). Time Point column will match those found in Section 8.9 of the SAP.

Maximum

XX

XX

XX

XX

P1R: < > P1M: < >

CIG: < >

Baseline is the last measurement collected prior to the first product administration.

Program: /CAXXXXX/sas prg/stsas/tab/programname2022Q1.sas DDMMYYYYY HH:MM

XX

XX


<sup># =</sup> Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

<sup>\* =</sup> Above reference range; ^ = Below reference range

# Philip Morris Products S.A. THS Induction device and regular or m

# THS Induction device and regular or menthol sticks, P1-PK-12 CA39924


Table CLBS Clinical Laboratory Shift From Baseline - Serum Chemistry (Safety Population)

| | | | Ba | selin | e L | Ba | selin | e N | Ba | seline | е Н |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Po | st Us | e | Po | st Us | e | Po | st Use | <br>e |
| Laboratory Test (units) | Randomized<br>Product Sequence | Time Point | <br>L | N | Н | L | N | Н | L | N | Н |
| Testname (unit) | XXX | Discharge | Х | XX | Х | X | XX | Х | X | XX | Х |
| | XXX | Discharge | X | XX | X | X | XX | X | X | XX | Χ |
| | XXX | Discharge | X | XX | X | X | XX | X | X | XX | Χ |
| | XXX | Discharge | X | XX | X | X | XX | X | X | XX | Χ |
| | XXX | Discharge | X | XX | X | X | XX | X | X | XX | Χ |
| | XXX | Discharge | X | XX | X | X | XX | X | X | XX | X |

Programmer Note: For urinalysis, the following footnote is used since the categories of N and O will be used instead of L, N, H: N = N within reference range; O = Outside reference range

P1R: < > P1M: < > CIG: < >

Baseline is the last measurement collected prior to the first product administration.

N = Within reference range; L = Below reference range; H = Above reference range


Table CVS Vital Sign Summary and Change From Baseline (Safety Population)

#### Randomized Product Sequence XXX XXX XXX XXX XXX XXX Vital Sign (units) Time Point (N = X)Statistic (N = X)(N = X)(N = X)(N = X)(N = X)Testname (unit) Baseline Χ Χ Χ Χ Χ Χ n Mean X.X X.X X.X X.X X.X X.X SD X.XX X.XX XXX.X X.XX XXX.X X.XX Minimum XX XX XX XX XX XX Median X.X X.X X.X X.X X.X X.X Maximum XXXX XXXXXX XXΧ Χ Χ Χ Χ Χ Day 2 Absolute n Mean X.X X.X X.X X.X X.X X.X SD X.XX X.XX X.XX X.XX X.XX X.XX Minimum XX XXXX XX XX XX Median X.X X.X X.X X.X X.X X.X Maximum XX XX XX XX XXXX Χ Χ Χ Χ Χ Χ Change n Mean X.X X.X X.X X.X X.X X.X SD X.XXX.XX X.XX X.XX X.XXX.XXMinimum XX XX XX XX XX XX Median X.X X.X X.X X.X X.X X.X

XX

XX

XX

XX

XX

XX

P1R: < > P1M: < > CIG: < >

Baseline is the last measurement collected prior to the first product administration.

Maximum


Table CEG 12-Lead Electrocardiogram Summary and Change From Baseline (Safety Population)

| | | | | | Rand | lomized Prod | luct Sequenc | e | |
|---|---|---|---|---|---|---|---|---|---|
| Measurement (units) | | | Statistic | (N = X) | (N = X) | (N = X) | (N = X) | (N = X) | (N = X) |
| Testname (unit) | | | n | Х | Х | Х | Х | Х | X |
| | | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |
| | Discharge | Absolute | n | X | X | X | X | X | X |
| | _ | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |
| | | Change | n | X | X | X | X | X | X |
| | | , | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |

P1R: < > P1M: < > CIG: < >

Baseline is the last measurement collected prior to the first product administration.

 $\label{program: program: pro$ 


Table CSP Spirometry Summary and Change From Baseline (Safety Population)

### Randomized Product Sequence

| Measurement (units) | Time Point | | Statistic | (N = X) $XXX$ | (N = X) | (N = X) | (N = X) | (N = X) | (N = X) |
|---|---|---|---|---|---|---|---|---|---|
| Testname (unit) | Baseline | | n | Х | X | X | X | Х | X |
| | | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |
| | Discharge | Absolute | n | Х | Х | X | Х | X | X |
| | _ | | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |
| | | Change | n | X | Х | X | X | X | X |
| | | - | Mean | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | SD | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | | | Minimum | XX | XX | XX | XX | XX | XX |
| | | | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | | | Maximum | XX | XX | XX | XX | XX | XX |

P1R: < > P1M: < > CIG: < >

Baseline is the last measurement collected prior to the first product administration .

### 13. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final report. Listings will generated from data created in accordance with SDTM Model 1.4 with Implementation Guide 3.2 or CDASH data structure. Listings with derived data may be created from the ADaM data. All listings will be presented in Courier New size font 9. Time point information (period, day, hour) will match that found in the CRF.

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges


| Laboratory Group | Test Name | Sex | Age Category | Reference Range | Unit |
|---|---|---|---|---|---|
| Serum Chemistry | Testname1<br>Testname2<br>ther tests, note that ag | MALE<br>MALE<br>e will only be pr | 0-25<br>26-99<br>resented when dif | XX - XXX<br>XX - XXX<br>XX - XXX<br>ferent reference ra | mEq/L<br>U/L<br>U/L<br>ange exists |
| Hematology | <similar che<="" serum="" td="" to=""><td>emistry&gt;</td><td></td><td></td><td></td></similar> | emistry> | | | |
| Urinalysis | Testname | MALE | | NEGATIVE | |
| Urine Drug Screening | Amphetamines | MAT.F. | | NOT DETECTED | |


### Appendix 16.2.1.1 Subject Disposition (Safety Population)

| | | Prematurely Discontinue From All Study Administration | | | | End of Study | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | 2 | Did Subject | | Primary Administra<br>Discontinuation<br>Reason | ation<br>Specify | Did Subject<br>Complete<br>the Study? | of Last | Primary Study<br>Discontinuation<br>Reason | Specify |
| 1<br>2 | XXX/XXX<br>XXX/XXX | No<br>No | | | | Yes<br>No | DDMMYYYY HH:MM<br>DDMMYYYY HH:MM | Personal Reason | xxxxx |
| 3 | XXX/X | Yes | DDMMYYYYY | Adverse Event | XXXXXXXXXXX | No | DDMMYYYYY HH:MM | Other | XXXXX |

P1R: THS regular stick P1M: THS menthol stick CIG: Combustible cigarette


### Appendix 16.2.1.2 Subject Disposition (Screen Failures)

#### End of Study

| Subject<br>Number | Did Subject<br>Complete<br>the Study? | Date of<br>Completion or<br>Discontinuation | Primary Study<br>Discontinuation<br>Reason | Specify |
|---|---|---|---|---|
| 1 | No<br>No | DDMMYYYY<br>DDMMYYYY | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| 3 | No | DDMMYYYY | Other | XXXXX |

P1R: THS regular stick P1M: THS menthol stick CIG: Combustible cigarette

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.4.2 will resemble the format of Appendix 16.2.4.1.

Appendix 16.2.4.1 Demographics (Safety Population)


| Subject<br>Number | Year Of<br>Birth | Age<br>(yr) | Sex | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | Body Mass<br>Index<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| 1 | YYYY<br>Similar to | 47 | Male | < > | Not Hispanic or Latino | XXX | XX.X | XX.XX |

# THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.4.4 will resemble the format of Appendix 16.2.4.3.

Appendix 16.2.4.3 Informed Consent (Safety Population)


| Subject<br>Number | | Informed | d Consent | In | Informed Re-consent | |
|---|---|---|---|---|---|---|
| | Date | Time | Protocol Version | Date | Time | Protocol Version |
| 1<br>2 | DDMMMYYYY<br><similar td="" to<=""><td>HH:MM<br/>above.</td><td>XXXXXXXXXXXX</td><td>DDMMYYYY</td><td>HH:MM</td><td>XXXXXXXXXXXX</td></similar> | HH:MM<br>above. | XXXXXXXXXXXX | DDMMYYYY | HH:MM | XXXXXXXXXXXX |
#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.4.6 will resemble the format of Appendix 16.2.4.5.

Appendix 16.2.4.5 Physical Examination (I of II) (Safety Population)

| Subject<br>Number | Study<br>Period | Date | Was Physical<br>Exam Performed? | System1 | System2 | System3 | System4 | System5 | System6 |
|---|---|---|---|---|---|---|---|---|---|
| X | Screen | DDMMMYY | YY Yes | NORMAL | NORMAL, | NORMAL, | NORMAL, | NORMAL, | NORMAL. |

<sup>\*</sup> = See Appendix 16.2.4.7 Physical Examination Description HEENT = Head, Eyes, Ears, Nose, Throat


Appendix 16.2.4.6 Physical Examination Descriptions (Safety Population)

| Subject<br>Number | | Date | System | Result | Description or Comment |
|---|---|---|---|---|---|
| | Screen | | Skin | ARNORMAT. | RICHT CHEST SCAR-NCS |

HEENT = Head, eyes, ears, nose, throat

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.4.8 Medical History (Safety Population)


| Subject | λnι | | | _ | Date | | |
|---|---|---|---|---|---|---|---|
| Number | History? | Condition or Event | System Organ Class | Preferred Term | Start | End | Ongoing? |
| 1 | No | | | | | | |
| 2 | Yes | < > | XXXXXXXX | xxxxxxxx | YYYY | | YES |

<note date can be YYYY, MONYYYY, or DDMONYYYY based on individual subject data>

Medical history are classified according to MedDRA Version 25.1.


Appendix 16.2.4.9 Tobacco/Nicotine-Containing Product Use History (Safety Population)

| Subject<br>Number | Study<br>Period | Was Assessment<br>Completed? | Date | Time | Product | Have You Smoked/Used<br>Continuously for at Least<br>the Past 3 Years? | In the Last 4 Weeks, on Average How Many of These Products did You Smoke/Use per Day? | |
|---|---|---|---|---|---|---|---|---|
| | Screen | XXX | DDMMMYYYY | HH•MM | XXXXXXX | XXX | XXXXXXXXXXXXXXX | _ |

CA39924

Appendix 16.2.4.10 Usual Brand Cigarettes Documentation (Safety Population)

| Page | ΩÍ |
|------|-----------------|
| Lage | <br>$O_{\perp}$ |

| Subject<br>Number | Study<br>Period | Substance | Start Date | Stop Date | Amount | Brand | Brand Style | Flavour | Cigarette Length |
|---|---|---|---|---|---|---|---|---|---|
| X | Screen | XXX | DDMMYYYY | DDMMYYYY | XXX | XXXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXXXX |

Appendix 16.2.4.11 Fagerström Test for Nicotine Dependence (Safety Population)

| | | | | | | | Quest | ion* | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Study<br>Period | Was Assessment Completed? | t<br>Date | Time | 1 2 3 4 5 6 | | | | | | <br>Total<br>Score | Classification of<br>Nicotine Dependence# |
| X | XXXX | XXX | DDMMMYYYY | HH:MM | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | <br>X | XXXXXXXXXX |

- \* 1 = .How soon after you wake up do you smoke your first cigarette?
- 2 = Do you find it difficult to refrain from smoking in places where it is prohibited?
- 3 = Which cigarette would you hate most to give up?
- 4 = How many cigarettes per day do you smoke?
- 5 = Do you smoke more frequently during the first hours after awakening than during the rest of the day?
- 6 = Do you smoke even if you are so sick that you are in bed most of the day?

#Classification score range: Mild (0 to 3 points); Moderate (4 to 6 points); Severe (7-10 points)

Program: /CAXXXXX/sas prg/stsas/lis/programname2022Q1.sas DDMONYYYY HH:MM


#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924


Appendix 16.2.5.1 Subject Enrollment (Safety Population) (Safety Population)

| Subject<br>Number | Study<br>Period | Study<br>Day | Was the Subject<br>Enrolled? | 21 | Criterion<br>ID Not Met | If Other, Specify |
|---|---|---|---|---|---|---|
| 1 | 1 | -X | YES | XXXXX | | |

### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.5.3 will resemble the format of Appendix 16.2.5.2.

 Appendix 16.2.5.2 Subject Eligibility (Safety Population)

| Subject<br>Number | Study<br>Period | Did subject meet all eligibility criteria? | Criterion<br>Not Met | Specify |
|---|---|---|---|---|
| 1 | Screen | YES | | |
| 2 | Screen | NO | Exclusion 5 | <pre><specify and="" be="" criterion="" if="" met="" not="" only="" populated="" presented="" will=""></specify></pre> |


Appendix 16.2.5.4 Randomization (Safety Population)

| Subject | Study | Study | Randomization | Randomization | Was the Subject | Randomization sequence |
|---|---|---|---|---|---|---|
| Number | Period | Day | Date | Time | Randomized? | |
| X | XXXX | XXX | DDMMYYYY | <br>HH:MM | XXXX | |

P1R: < > P1M: < > CIG: < >


Appendix 16.2.5.5 Investigational Product Administration (Safety Population)

| | | | | | | Product Use | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Study | | | | | | | Planned Product | |
| Number | Period | Product | Day | Interval | Date | Start Time | Stop Time | and Unit | Comments |
| 1 | 1 | XXX | 1 | XX-XX | DDMMYYYYY | HH:MM:SS | HH:MM:SS | XXXXXXXX | XXXXXXXX |

P1R: < > P1M: < > CIG: < >

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

#### Appendix 16.2.5.6 Prior and Concomitant Medications (Safety Population)

| Subject<br>Number | Product | Prior? | Medication<br>(WHO DD) | Dosage | Route | Start<br>Date | Start<br>Time | End<br>Date | End<br>Time | Frequency | Indication | Ongoing? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | | | None | | | | | | | | | |
| 2 | | | None | | | | | | | | | |
| 3 | | Yes | CETIRIZINE<br>(CETIRIZINE) | X MG | BY MOUTH | DDMONYYYY | | DDMONYYYY | HH:MM | XXXXXX | XXXXXXX | NO |
| | XXX | No | PARACETAMOL<br>(PARACETAMOL) | X MG | XXXXXXXX | DDMONYYYY | HH:MM | XXXXXXXX | HH:MM | XXXXXXX | XXXXXXX | XX |

P1R: < > P1M: < > CIG: < >

Concomitant medications are coded with WHO Drug Dictionary Version 01SEP2022 b3.

WHO DD = World Health Organization Drug Dictionary

Prior is defined as a medication administered prior to the first study product administration.

Program: /CAXXXXX/sas prg/stsas/lis/programname2022Q1.sas DDMONYYYY HH:MM


Appendix 16.2.5.7 Plasma Nicotine Pharmacokinetic Blood Draw Times and Concentration Data (Safety Population)

| Subject | Period | Study | | CRF | Blood | Draw | Elapsed<br>Time From<br>Last Product Use | Measured<br>Concentration | |
|---|---|---|---|---|---|---|---|---|---|
| Number | | | Day | Timepoint | Date | Time | (minutes) | (ng/mL) | Comment |
| 1 | 1 | P1R | 1 | XXXXX | DDMONYYYY<br>DDMONYYYY | HH:MM:SS<br>HH:MM:SS | 0.00<br>X.XX | x.xx<br>x.xx | |
| | | | < > | XXXXX<br>> | DDMONYYYY | HH:MM:SS | X.XX | X.XX | |

<similar for all other time points and subjects>

P1R: < > P1M: < > CIG: < >

Program: /CAXXXX/sas\_prg/pksas/standardlis/pk\_bld.sas DDMMYYYY HH:MM Programmer Notes:

• Population: Safety population will be used in this listing.

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.6.2 VAS Craving Assessment (Safety Population)


| Subject<br>Number | Study<br>Period | Study<br>Product | Study<br>Day | Study<br>Hour | Date | Was Event<br>Performed? | VAS Score | Comment | |
|---|---|---|---|---|---|---|---|---|---|
| X | X | XXX | XXXX | X.XX | DMMMYYYY | XXX | XXX | | <br> |

P1R: < > P1M: < > CIG: < >

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.6.3 VAS Liking Assessment (Safety Population)


| Subject<br>Number | Study<br>Period | Study<br>Product | Study<br>Day | Study<br>Hour | Date | Was Event<br>Performed? | VAS Score | Comment |
|---|---|---|---|---|---|---|---|---|
| X | X | XXX | XXXX | X.XX | DMMYYYY | XXX | XXX | |

P1R: < > P1M: < > CIG: < >

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.6.4 Intention to Use Again (Safety Population)


| Subject<br>Number | Study<br>Period | Study<br>Product | Study<br>Day | Study<br>Hour | Date | Was Event<br>Performed? | VAS Score | Comment |
|---|---|---|---|---|---|---|---|---|
| X | Х | XXX | XXXX | X.XX | DMMYYYY | XXX | XXX | |

P1R: < > P1M: < > CIG: < >

#### THS Induction device and regular or menthol sticks, P1-PK-12

#### CA39924

#### Appendix 16.2.7.1 Adverse Events (Safety Population)

| rage |
|------|

| Subject<br>Number | Age/<br>Sex | Product | PUE? | System Organ Class/<br>Preferred Term<br>(Verbatim) | Time From<br>Last Use<br>(DD:HH:MM) | Date:Time<br>End<br>Duration | , | Serious/<br>Outcome | Severity/<br>Frequency | Study Product<br>Relationship/<br>Action/<br>Other Action | Study Procedure<br>Relationship/<br>Expectedness |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 30/F | | | None | | | | | | | |
| 2 | 24/M | | | None | | | | | | | |
| 3 | 52/M | XXX | | XXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXX | | DDMONYYYY:F<br>DDMONYYYY:F<br>00:23:15 | | No/<br>Recovered/<br>Resolved | Moderate/<br>Intermittent | Related/<br>XXXXXXX/<br>XXXXXXXXXX | Unrelated/<br>Expected |
| | | XXX | Yes | <similar above="" to=""></similar> | | | | | | | |
| 4 | XX/M | SFU | Yes | XXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXX | | DDMONYYYY:FDDMONYYYY:F00:23:15 | | No/<br>Recovered/<br>Resolved | Moderate/<br>Intermittent | Related/<br>XXXXXXX/<br>XXXXXXXXXX | Unrelated/<br>Expected |

Programmer Note: AEs should be presented start date/time order for each subject.

P1R: < > P1M: < >

CIG: < >

Adverse events are classified according to MedDRA Version 25.1

PUE = Abbreviation for product use-emergent

F = Female; M = Male

SFU = after discharge from CRU to safety follow-up visit

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924


Appendix 16.2.7.2 Details for Serious Adverse Events (Safety Population)

Persistent or

| Subject<br>Number | | | | System Organ Class/<br>Preferred Term<br>(Verbatim) | End | Serious | Anomaly/ | Significant<br>Disability or<br>Incapacity? | _ | | | Death? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 3 | 52/M | P1R | Yes | | DDMONYYYY<br>DDMONYYYY<br>00:23:15 | Yes | No | No | Yes | No | Yes: < > | No |

Programmer Note: If Serious = Yes then present AEs in this listing otherwise please do not include this listing.

P1R: < > P1M: < > CIG: < >

Adverse events are classified according to MedDRA Version 25.1.

PUE = Abbreviation for product use-emergent

F = Female; M = Male

SFU = after discharge from CRU to safety follow-up visit

CA39924


Appendix 16.2.7.3 Product Events (Safety Population) (Safety Population)

| Subject<br>Number | J . | roduct | Any<br>Events? | Date | Time | Device<br>Number | Affected<br>Part | Severity | Event<br>Category | Description of<br>Product Event/<br>Complaint | Was Pharmacy<br>Informed? | | New Device<br>Serial<br>Number |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 3 | 52/M | P1R | <br>Yes | DDMMYYYY | HH:MM:SS | XXXX | XXXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXXX |

P1R: < > P1M: < > CIG: < >

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

#### Appendices 16.2.8.2 – 16.2.8.5 will resemble 16.2.8.1.

Appendix 16.2.8.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)


| Subject<br>Number | | Study<br>Period | Day | Hour | Date | Time | Chloride<br>M: 97-105<br>(mEq/L) | Potassium<br>M: 3.7-5.2<br>(mEq/L) | Phosphorus<br>M: 2.4-4.4<br>(mg/dL) | Sodium<br>M: 135-143<br>(mEq/L) |
|---|---|---|---|---|---|---|---|---|---|---|
| 1 | XX/M | Screen<br>1<br>Recheck | 1 | -17.00 | DDMONYYYY<br>DDMONYYYY<br>DDMONYYYY | HH:MM:SS | XXX<br>XXX HN<br>XXX | X.X<br>X.X<br>X.X | X.X<br>X.X<br>X.X | XXX HY- G1<br>XXX HN<br>XXX |

<similar to above for all subjects/time points>

```
F = Female; M = Male

H = Above reference range

CS flag: N = Not clinically significant; Y = Clinically significant

PI interpretation: - = Not clinically significant

CTCAE grade (Version 5.0): G1 = Mild
```


Appendix 16.2.8.6 Alcohol Breath Test (Safety Population)

| Subject<br>Number | | | Date | Time | Result | & Unit | Comment |
|---|---|---|---|---|---|---|---|
| 1 | XX/M | Screen | DDMONYYYY H | H:MM:SS | XXX | XXX | |

<similar to above for all subjects/time points>

F = Female; M = Male

### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

Appendix 16.2.8.7 Vital Signs (Safety Population)


| | | | | | | | | d Pre<br>(mmHg | ssure<br>() | | Respir- | Temper- | - |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | | | Day | Hour | Date | Time | Position | <br>n | Sys/Dia | Pulse<br>(bpm) | | ature<br>(°C) | Weight<br>(kg) |
| 1 | 30/F | Screen | | | DDMONYYYY | HH:MM:SS | SUP5 | XXX/ | | · | xx xx | | XX.X |
| | | | | | R<br>R | HH:MM:SS<br>HH:MM:SS | SUP5 | XXX/ | XX | 21 . | 701 701 | • 21 | |
| | | 1 | -1 | -17.0 | DDMONYYYY | | | XXX/ | | | | | |

F = Female; M = Male SUP5 = 5-minute supine; R = Recheck value; brpm = breaths/min

### THS Induction device and regular or menthol sticks, P1-PK-12 CA39924

Appendix 16.2.8.8 12-Lead Electrocardiogram (Safety Population)


| | | Study<br>Period | Day | Hour | Date | Time | Result | Heart<br>Rate<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF<br>(msec) | Specify/Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 30/F | Screen | | | DDMONYYYY | X:XX:XX | WNL | XX | XX | XX | XXX | XXX | EARLY REPOLARIZATION;<br>LEFT AXIS DEVIATION |
| | | 1 3 | _ | X.XX<br>X.XX | | XX:XX:XX<br>XX:XX:XX | ANCS<br>< > | XX<br>XX | XX<br>XX | XX<br>XX | XXX | 410<br>451 | LEFT AXIS DEVIATION SINUS BRADYCARDIA |

F = Female; M = Male

 $R = Recheck\ value;\ WNL = Within\ normal\ limits;\ ANCS = Abnormal,\ not\ clinically\ significant\ QTcF = QT\ corrected\ for\ heart\ rate\ using\ Fridericia's\ correction$ 

#### THS Induction device and regular or menthol sticks, P1-PK-12

CA39924

#### Appendix 16.2.8.9 Spirometry (Safety Population)


| | | Study<br>Period I | Day | Hour | Date | Time | / | FVC<br>Predicted<br>(%) | FEV1<br>(L) | FEV1<br>Predicted<br>(%) | FEV1/FVC<br>Ratio | Abnormal? | If Abnormal,<br>Indicate if<br>CS/NCS | Comment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 30/F | Screen<br>1 | Х | | DDMONYYYY<br>DDMONYYYY | | | | XX<br>XX | XXX<br>XXX | XXX<br>XXX | X<br>X | | |

F = Female; M = Male

NCS = Not clinically significant; CS = Clinically significant 15? = Did subject rest for at least 15 minutes in sitting position?

1h? = Did subject not use cigarettes for at least 1 hour?